CLINICAL TRIAL: NCT00346216
Title: A Randomized, Double Blind, Parallel-group Study Of Cardiovascular Safety In Osteoarthritis Or Rheumatoid Arthritis Patients With Or At High Risk For Cardiovascular Disease Comparing Celecoxib With Naproxen And Ibuprofen
Brief Title: Prospective Randomized Evaluation Of Celecoxib Integrated Safety Vs Ibuprofen Or Naproxen
Acronym: PRECISION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A3191172; 2004-002441-13 (EudraCT Number); PRECISION TRIAL (Other: Alias Study Number)
Record Dates: First submitted 2006-06-28; First posted 2006-06-29 (Estimated); Results first posted 2017-05-01 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Celecoxib; Ibuprofen; Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- celecoxib (Experimental): subject receives celecoxib and dummy (placebo) ibuprofen and naproxen
  Interventions: Drug: celecoxib
- ibuprofen (Active Comparator): subject receives ibuprofen and dummy (placebo) celecoxib and naproxen
  Interventions: Drug: Ibuprofen
- naproxen (Active Comparator): subject receives naproxen and dummy (placebo) celecoxib and ibuprofen
  Interventions: Drug: Naproxen

INTERVENTIONS:
Drug: celecoxib — 100 to 200 mg twice daily, taken by mouth
  Arms: celecoxib
Drug: Ibuprofen — ibuprofen 600 mg to 800 mg three times daily, taken by mouth
  Arms: ibuprofen
Drug: Naproxen — naproxen 375mg to 500 mg twice daily, taken by mouth
  Arms: naproxen

SUMMARY:
To answer the question of overall benefit: risk of celecoxib when compared to two most commonly prescribe traditional (non-selective) nonsteroidal anti-inflammatory drugs (NSAIDs) in the treatment of arthritis pain. For this purpose, patients with osteoarthritis or rheumatoid arthritis with or at risk of developing cardiovascular disease will be recruited. The cardiovascular, gastrointestinal and renal safety and symptomatic benefit in each treatment group will be assessed accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with osteoarthritis or rheumatoid Arthritis with or at risk of developing cardiovascular disease and who require and eligible for chronic, daily therapy with an NSAID to control arthritis sign and symptoms.

Exclusion Criteria:

* Subjects have had a recent cardiovascular event, unstable cardiovascular conditions, or any major surgery (cardiac or non-cardiac) within 3 months prior to randomization;
* Subjects with medical or laboratory abnormality that would make the subject inappropriate for entry into this trial
* Subjects require treatment with aspirin > 325 mg /day
* Subjects with known hypersensitivity to celecoxib, ibuprofen, naproxen, aspirin or esomeprazole, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24081 (Actual)
Dates: Start 2006-10-04 (Actual); Primary Completion 2016-04-12 (Actual); Study Completion 2016-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1061):
- United States (866):
  - Carol M. Johnson MD, LLC, Alabaster, Alabama
  - Orthopaedics West, Bessemer, Alabama
  - Central Alabama Research, Birmingham, Alabama
  - Simon Williamson Clinic/Clinical Research Advantage, Inc., Birmingham, Alabama
  - Achieve Clinical Research, LLC, Birmingham, Alabama
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - Cahaba Research Inc., Birmingham, Alabama
  - Winston Technology Inc., Haleyville, Alabama
  - Clinical Research Consultants, Inc, Hoover, Alabama
  - Medical Affiliated Research Center, Incorporated, Huntsville, Alabama
  - Rheumatology Associates of North Alabama, PC, Huntsville, Alabama
  - Montgomery Rheumatology Associates, Montgomery, Alabama
  - James P. Beretta, PC, Pelham, Alabama
  - Alabama Clinical Research Associates, Pell City, Alabama
  - Pell City Internal and Family Medicine, Pell City, Alabama
  - Scottsboro Quick Care Clinic, Scottsboro, Alabama
  - Clinic for Rheumatic Diseases, Tuscaloosa, Alabama
  - Terence T. Hart , MD, Tuscumbia, Alabama
  - Clinical Research Advantage Inc./ Warner Family Practice, PC, Chandler, Arizona
  - ArthroCare, Arthritis Care & Research P.C., Gilbert, Arizona
  - Clinical Research Advantage Inc., /Thunderbird Internal Medicine, Glendale, Arizona
  - Arizona Center for Clinical Research, Glendale, Arizona
  - Clinical Research Advantage, Inc./ Lenzmeier Family Medicine, Glendale, Arizona
  - Clinical Research Advantage, Inc./Central Arizona Medical Associates, PC, Mesa, Arizona
  - Novara Clinical Research, Mesa, Arizona
  - Clinical Research Advantage, Inc., Mesa, Arizona
  - Sun Valley Arthritis Center, Limited, Peoria, Arizona
  - Lovelace Scientific Resources, Inc., Phoenix, Arizona
  - Clinical Research Advantage, Inc./ Family Practice Specialists, LTD, Phoenix, Arizona
  - NPHC Research, Phoenix, Arizona
  - Phoenix Clinical, Phoenix, Arizona
  - Arizona Research Center, Inc., Phoenix, Arizona
  - Precision Trials AZ. LLC; AZ, Phoenix, Arizona
  - 43rd Medical Associates, P.C., Phoenix, Arizona
  - Southwest Health Ltd., Scottsdale, Arizona
  - Advanced Arthritis Care and Research, Scottsdale, Arizona
  - Arizona Pain Specialist, PLLC, Scottsdale, Arizona
  - Sonora Quest Laboratories, Scottsdale, Arizona
  - Cochise Clinical Research, Sierra Vista, Arizona
  - Clinical Research Advantage, Inc./Skyline Medical Center PC, Tempe, Arizona
  - Clinical Research Advantage, Inc./Urban Family Practice Associates, PC, Tempe, Arizona
  - Clinical Research Advantage, Inc./Warner Family Practice, PC, Tempe, Arizona
  - Clinical Research Advantage, Inc/Manning Family Care, Tempe, Arizona
  - Clinical Research Advantage, Incl Colorado Springs Health Partners, East, Tempe, Arizona
  - Family Medicine Associates/Clinical Research Advantage, Tempe, Arizona
  - Clinical Research Advantage, Inc./Fiel Family and Sports Medicine, PC, Tempe, Arizona
  - ARA-Arizona Research Associates, Tucson, Arizona
  - Canyon Clinical Research LLC, Tucson, Arizona
  - Tucson Clinical Researh, Tucson, Arizona
  - ACRC/Arizona Clinical Research Center, Incorporated, Tucson, Arizona
  - Clinical Research Advantage, Inc./ Orange Grove Family Practice, Tucson, Arizona
  - Genova Clinical Research, Tucson, Arizona
  - Eclipse Clinical Research, Tucson, Arizona
  - Fayetteville Diagnostic Clinic Limited, Fayetteville, Arkansas
  - Hearne Family Practice Clinic, Little Rock, Arkansas
  - Larry S. Watkins, M.D., Little Rock, Arkansas
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - Rx Medical Research of AR, Little Rock, Arkansas
  - Anaheim Family Medical Center, Anaheim, California
  - Advanced Research Center, Anaheim, California
  - Advanced Arthritis & Rheumatology Center, Artesia, California
  - Bina Akamdar MD, Azusa, California
  - Rx for Life, Inc, Bell, California
  - Clinical Research Advantage Inc., /Cassidy Medical Group-Carlsbad, Carlsbad, California
  - Capitol Interventional Cardiology, Carmichael, California
  - Northern California Research, Carmichael, California
  - CORE Orthopaedic Medical Center, Encinitas, California
  - Arthritis Medical Clinic of North County, Inc., Escondido, California
  - Med Investigations, Inc., Fair Oaks, California
  - Valley Research, Fresno, California
  - Creekside Clinical Research, Greenbrae, California
  - C. V. Mehta, MD Medical Corporation, Hemet, California
  - Talbert Medical Group, Huntington Beach, California
  - Alia Clinical Research, Inc, Huntington Park, California
  - Time Clinical Research Inc., Huntington Park, California
  - Lindora Research Center, Irvine, California
  - Office of Dr. Robert L. Freed, MD, Irvine, California
  - Office of Dr. Alan Schenk, Laguna Hills, California
  - Prime Care Clinical Research, Laguna Hills, California
  - Jeremy Anuntiyo, Lakewood, California
  - Premiere Clinical Research, LLC, Lakewood, California
  - Stuart J. Finkelstein, Lakewood, California
  - Clinical Trials Research, Lincoln, California
  - VA Loma Linda Healthcare System, Loma Linda, California
  - Narbonne Multi-Specialty Medical Group Inc., Lomita, California
  - Office of Dr. Arvind J. Mehta, Long Beach, California
  - Pacific Internal Medicine Group, Inc, Long Beach, California
  - Long Beach Center for Clinical Research, Long Beach, California
  - National Institute of Clinical Research, Long Beach, California
  - Alliance Research, LLC, Long Beach, California
  - Valerius Medical Group and Research Center, Los Alamitos, California
  - IMD Medical Group, Los Angeles, California
  - Pacific Arthritis Care Center, Los Angeles, California
  - Wagdy W. Kades, MD, Inc., Los Angeles, California
  - Samaritan Center for Medical Research Medical Group, Los Gatos, California
  - Office of Lewis Gamarra, MD M.P.H., Los Osos, California
  - Adegbenga A. Adetola, M.D., Lynwood, California
  - Facey Medical Group, Mission Hills, California
  - Providence Clinical Research, North Hollywood, California
  - Desert Medical Group, Palm Springs, California
  - The Office of Dr. Marcos Yang, Palos Verdes Estates, California
  - Bayview Research Group, LLC, Paramount, California
  - Sierra Rheumatology, Roseville, California
  - Center for Clinical Trials of Sacramento, Inc., Sacramento, California
  - Sacramento Heart and Vascular Research Center, Sacramento, California
  - California Research Foundation, San Diego, California
  - San Diego Arthritis Medical Clinic, San Diego, California
  - Wetlin Research Associates, Inc, San Diego, California
  - Medical Associates Research Group, San Diego, California
  - San Jose Valley Research, Inc., San Jose, California
  - Comprehensive Adult Risk Evaluation, San Leandro, California
  - East Bay Rheumatology Medical Group Inc, San Leandro, California
  - Central Coast Pathology Consultants, San Luis Obispo, California
  - Coastal Medical Research Group, Inc., San Luis Obispo, California
  - Family Medical Center, San Luis Obispo, California
  - Office of Ajay G. Meka, MD, Santa Ana, California
  - Pacific Arthritis Center Medical Group, Santa Maria, California
  - Orrin M. Troum & Medical Associates, Santa Monica, California
  - Northern California Medical Associates, Santa Rosa, California
  - Robert Simon, MD, Sherman Oaks, California
  - St. Joseph Medical Associates, Stockton, California
  - Westlake Medical Research, Thousand Oaks, California
  - Paradigm Clinical Research Institute, Inc., Torrance, California
  - Orange County Research Center, Tustin, California
  - Inland Rheumatology and Osteoporosis Medical Group, Upland, California
  - Inland Rheumatology Clinical Trials, Inc., Upland, California
  - Bayview Research Group, Valley Village, California
  - Medvin Clinical Research, Van Nuys, California
  - Center for Clinical Trials of San Gabriel, West Covina, California
  - Agilence Arthritis and Osteoporosis Medical Center, Inc., Whittier, California
  - Avalon Family Medical Group, Wilmington, California
  - Darrell E. Gorman, MD, Arvada, Colorado
  - Aurora Denver Cardiology Associates, Aurora, Colorado
  - Azmi Emil Farag, MD, Colorado Springs, Colorado
  - Lynn Institute of the Rockies, Colorado Springs, Colorado
  - Colorado Springs Health Partners- East/Clinical Research Advantage, Colorado Springs, Colorado
  - Mountain View Clinical Research, Inc., Denver, Colorado
  - Saint Luke's Medical Clinic, Fort Collins, Colorado
  - New West Physicians, Golden, Colorado
  - Ranch View Family Medicine, Highlands Ranch, Colorado
  - Colorado Center for Bone Research PC, Lakewood, Colorado
  - South Denver Cardiology Associates, PC, Littleton, Colorado
  - Lynn Institute of Pueblo, Pueblo, Colorado
  - Connecticut Clinical Research, LLC, Bridgeport, Connecticut
  - Connecticut Gastroenterology Institute, Bristol, Connecticut
  - Arthritis and Osteoporosis Center, PC, Hamden, Connecticut
  - Robert Lang, MD, P.C., Hamden, Connecticut
  - Coastal Connecticut Research, LLC, New London, Connecticut
  - Office of Edward J. McDermott, Jr., MD, New London, Connecticut
  - Orthopaedics Foundation for Active Lifestyles, Stamford, Connecticut
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - New England Research Associates, LLC, Trumbull, Connecticut
  - Arthritis Center of Connecticut, Waterbury, Connecticut
  - Rheumatology Consultants of Delaware, Lewes, Delaware
  - Office of Cynthia Morgan, MD, Washington D.C., District of Columbia
  - The Center for Rheumatology and Bone Research, Washington D.C., District of Columbia
  - Medical Specialist of the Palm Beaches, Atlantis, Florida
  - South Florida Medical Research, Aventura, Florida
  - RASF - Clinical Research Center, Boca Raton, Florida
  - Orthopedic Research Institute, Boynton Beach, Florida
  - Clinical Research of Brandon, LLC, Brandon, Florida
  - Family Healthcare of Chipley, Chipley, Florida
  - Health First Clinical Research Group, Inc., Chipley, Florida
  - Southern Family Healthcare and Health First Research Group Inc., Chipley, Florida
  - Florida Research & Testing, LLC, Clearwater, Florida
  - Alba Clinical Research, Clearwater, Florida
  - Appletree Medical, Clearwater, Florida
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - Clinical Research of West Florida, Clearwater, Florida
  - Rameshwar N. Mathur, MD, PA, Cocoa, Florida
  - Nature Coast Clinical Research, LLC, Crystal River, Florida
  - Atlantic Institute of Clinical Research, Daytona Beach, Florida
  - International Medical Research, Daytona Beach, Florida
  - Omega Research Consultants, LLC, DeBary, Florida
  - Physicians Research Alliance, LLC, DeBary, Florida
  - Deerfield Beach Cardiology Associates, Deerfield Beach, Florida
  - Doctors Medical Center of Walton County, DeFuniak Springs, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - Florida Research Associates, LLC/Florida Orthopaedic Associates, P.A., DeLand, Florida
  - Cohen Medical Associates, PA, Delray Beach, Florida
  - Clark Family Medicine & Emerald Coast Research Group, Destin, Florida
  - SJS Clinical Research, Inc, Destin, Florida
  - Robert W. Levin MD, Dunedin, Florida
  - Riverside Clinical Research, Edgewater, Florida
  - Fleming Island Center for Clinical Research, Fleming Island, Florida
  - Invesclinic, Fort Lauderdale, Florida
  - M&O Clinical Research, LLC, Fort Lauderdale, Florida
  - Maxine Hamilton, MD PA, Fort Lauderdale, Florida
  - Holy Cross Medical Group Northridge Internal Medicine, Fort Lauderdale, Florida
  - Clinical Physiology Associates, Fort Myers, Florida
  - Emerald Coast Mood & Memory, Fort Walton Beach, Florida
  - White-Wilson Medical Center, PA, Fort Walton Beach, Florida
  - Cardiology West, Gainesville, Florida
  - Florida Research Network, LLC, Gainesville, Florida
  - Southeastern Integrated Medical, PL, Gainesville, Florida
  - Shands at the University of Florida, Gainesville, Florida
  - University of Florida, Gainesville, Florida
  - Genetic Medical Research Corporation, Hialeah, Florida
  - Direct Helpers Medical Center, Inc., Hialeah, Florida
  - Indago Research & Health Center, Inc., Hialeah, Florida
  - Reliable Clinical Research, LLC, Hialeah, Florida
  - Orthopaedic Associates of South Broward, P.A., Hollywood, Florida
  - Advanced Research Institute of Miami, Homestead, Florida
  - Pasco Cardiology Center, Hudson, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - Westside Center for Clinical Research, Jacksonville, Florida
  - East Coast Institute for Research, LLC, Jacksonville, Florida
  - Jacksonville Center for Clincal Research, Jacksonville, Florida
  - St. Vincent's Cardiology, Jacksonville, Florida
  - Dr. Ricardo A. Bedoya, M.D., Jupiter, Florida
  - Drug Study Institute, Jupiter, Florida
  - Christopher Chappel, Kissimmee, Florida
  - Florida Arthritis Center, LLC, Lake Mary, Florida
  - Pedro Ylisastigui, MD, Lehigh Acres, Florida
  - Adult Medicine Specialists, Longwood, Florida
  - Genesis Research International, Longwood, Florida
  - Doctors Inn, Madeira Beach, Florida
  - Everest Medical Care and Palm Court Research Group, Marianna, Florida
  - Panhandle Family Care Associates & Emerald Coast Research Group, Marianna, Florida
  - The Doctor's Office, Marianna, Florida
  - Health First Medical Group, Melbourne, Florida
  - Holmes Regional Medical Center, Melbourne, Florida
  - Pharmaceutical Research Associates, Merritt Island, Florida
  - Homestead Associates in Research, Inc, Miami, Florida
  - Pharmax Research Clinic, Miami, Florida
  - Life Spring Research Foundation, Miami, Florida
  - Miami International Cardiology Consultants, Miami, Florida
  - Florida Medical Center & Research, Inc., Miami, Florida
  - The Center for Arthritis and Rheumatic Diseases, Miami, Florida
  - Well Pharma Medical Research Corporation, Miami, Florida
  - DC Health Clinical Trials, Miami, Florida
  - School of Clinical Research USA, LLC, Miami, Florida
  - Advance Medical Research Services, Corp, Miami, Florida
  - Future Care Solution, LLC, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Miami Cardiology Group, Miami, Florida
  - M & M Medical Center, Miami, Florida
  - Office of Dr. Juvenal E. Martinez, MD, PA, Miami, Florida
  - Orthopaedic Specialist of Miami Beach, Miami Beach, Florida
  - AMPM Research Clinic, Miami Gardens, Florida
  - Crystal Biomedical Research, LLC, Miami Lakes, Florida
  - Pembroke Clinical Trials, Miami Lakes, Florida
  - Anchor Research Center, Naples, Florida
  - Jeffrey Alper M.D. Research, Naples, Florida
  - Anchor Health Centers, Naples, Florida
  - Medical Surgical Specialists, Physicians Regional Medical Center, Naples, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Magnolia Research Group, Inc., Ocala, Florida
  - Ocala Rheumatology Research Center, Ocala, Florida
  - Paddock Park Clinical Research, Ocala, Florida
  - Southeastern Rehabilitation Medicine, Ocala, Florida
  - Tequesta Research Group, Ocala, Florida
  - CEC Research, INC., Ocoee, Florida
  - Florida Heart Group, PA, Orlando, Florida
  - Florida Hospital, Orlando, Florida
  - Compass Research, LLC, Orlando, Florida
  - DCT FMC, LLC dba Discovery Clinical Trials, Orlando, Florida
  - DCT-FMC, LLC dba Discovery Clinical Trials, Orlando, Florida
  - Arthur L. Hall MD PA, Orlando, Florida
  - Block and Nation, PA, Oviedo, Florida
  - Arthritis Research of Florida, Inc., Palm Harbor, Florida
  - Florida Med Center of Countryside, Palm Harbor, Florida
  - Rene CaSanova Medical Office Inc, Pembroke Pines, Florida
  - Boulevard Professional Centre, Pembroke Pines, Florida
  - Research Physician Network Alliance, Pembroke Pines, Florida
  - South Broward Research LLC, Pembroke Pines, Florida
  - South Florida Research Solutions, LLC, Pembroke Pines, Florida
  - DMI Research, Inc., Pinellas Park, Florida
  - Sunbelt Research, LLC, Plantation, Florida
  - Boca Raton Clinical Research, Plantation, Florida
  - St. Johns Center for Clinical Research, Ponte Vedra, Florida
  - Accord Clinical Research, LLC, Port Orange, Florida
  - Administrative Address: Florida Arthritis & Osteoporosis Center, Port Richey, Florida
  - Heart & Vascular Center Research, Sarasota, Florida
  - Edgar R. Blecker, MD, Sebastian, Florida
  - Phoenix Clinical Research, LLC., Tamarac, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - Soutwest Florida Clinical Research Center, Tampa, Florida
  - Clinyx/Floria Cardiovascular, Tampa, Florida
  - Stedman Clinical Trials, LLC, Tampa, Florida
  - West Wind'r Research, Tampa, Florida
  - Health Point Medical Group, Inc, Tampa, Florida
  - Causeway Medical Clinic, Tampa, Florida
  - Office of Alastair C. Kennedy, MD, Vero Beach, Florida
  - Metabolic Research Institute, Incorporated, West Palm Beach, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Central Florida Primary Care, Winter Park, Florida
  - Florida Medical Clinic, PA, Zephyrhills, Florida
  - The Kaufmann Clinic, Atlanta, Georgia
  - Piedmont Heart Institute, Atlanta, Georgia
  - Arthritis and Rheumatology of Georgia, Atlanta, Georgia
  - Atlanta Center for Clinical Research, Corp., Atlanta, Georgia
  - Atlanta Vascular Research Foundation, Atlanta, Georgia
  - Executive Health and Research Associates, Atlanta, Georgia
  - Southern Clinical Research and Management, Inc. (SCRAM), Augusta, Georgia
  - Masters of Clinical Research, Inc., Augusta, Georgia
  - Amelia Medical Plaza, Bainbridge, Georgia
  - Bainbridge Medical Associates, Bainbridge, Georgia
  - Abdul Bari MD Inc, Cairo, Georgia
  - Southern Clinical Research Management and Consulting, Cairo, Georgia
  - North Georgia Rheumatology Group, PC, Duluth, Georgia
  - United Osteoporosis Centers, Gainesville, Georgia
  - North Georgia Rheumatology Group, PC, Lawrenceville, Georgia
  - GCH Research Dr. G Craig Heigerick DO, Lilburn, Georgia
  - Mercer University Mercer Medicine, Macon, Georgia
  - Drug Studies America, Marietta, Georgia
  - Clinical Research Advantage, Inc./Urban Family Practice Associates, PC, Marietta, Georgia
  - In-Quest Medical Research, LLC, Norcross, Georgia
  - Harbin Clinic, Rome, Georgia
  - Atlanta Center for Clinical Research, Roswell, Georgia
  - Herman Clinical Research, LLC, Suwanee, Georgia
  - Archibold Primary Care, Thomasville, Georgia
  - Clinical Trial Providers, Inc., Tucker, Georgia
  - VSC, Valdosta, Georgia
  - Kaufmann Clinic, INC, Woodstock, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - North Georgia Internal Medicine, Woodstock, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Orthopedic Health Care Clinic, Boise, Idaho
  - Sonora Clinical Research, LLC, Boise, Idaho
  - Eagle's View Family Medicine, Boise, Idaho
  - Coeur D'Alene Arthritis Clinic, Coeur d'Alene, Idaho
  - CTL Research, Eagle, Idaho
  - Women's Healthcare Associates P.A. dba Rosemark WomenCare Specialists, Idaho Falls, Idaho
  - Idaho Arthritis and Osteoporosis Center, Meridian, Idaho
  - Advanced Clinical Research, Meridian, Idaho
  - AMR Sakeena Research, Aurora, Illinois
  - Arthur I Davida, MD PC, Bloomingdale, Illinois
  - Cardiac Wellness Consultants, Chicago, Illinois
  - Chicago Peripheral Nerve Center, Chicago, Illinois
  - ICCT Research International Incorporated, Chicago, Illinois
  - Claude Mandel Medical Center, Chicago, Illinois
  - Windy City Orthopedics and Sports Medicine, Evanston, Illinois
  - South Suburban Health Professional Group, Hazel Crest, Illinois
  - Prairie Rheumatology Associates, SC, Joliet, Illinois
  - Lake Zurich Family Treatment Center, Lake Zurich, Illinois
  - Southern Illiniois Clinical Research Centre, O'Fallon, Illinois
  - Speciality phhysicians of Illinois, LLC, Olympia Fields, Illinois
  - Redhead Research Inc., DBA Research Associates of Central Illinois, Peoria, Illinois
  - Trinity Medical Center, Rock Island, Illinois
  - Rockford Health Physicians, Rockford, Illinois
  - Prairie Cardiovascular Consultants, Springfield, Illinois
  - Prairie Education & Research, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Deerbrook Medical Associates, Vernon Hills, Illinois
  - Community Clinical Research Center, Anderson, Indiana
  - American Health Network of Indiana, LLC, Avon, Indiana
  - Robert D. Barnes, MD, LLC, Evansville, Indiana
  - Clinical Research Advantage, Inc., Evansville, Indiana
  - Destiny Clinical Research, LLC, Evansville, Indiana
  - Clinical Research Advantage/Family Medicine Associates, Evansville, Indiana
  - American Health Network of Indiana, LLC, Franklin, Indiana
  - Internal Medicine Center of Northwest Indiana, P.C., Gary, Indiana
  - Beacon Medical Group Rheumatology, Granger, Indiana
  - American Health Network of IN, LLC, Greenfield, Indiana
  - Diagnostic Rheumatology And Research, PC, Indianapolis, Indiana
  - Investigators research Group, Indianapolis, Indiana
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Dawes Fretzin Dermatology Group, LLC, Indianapolis, Indiana
  - Arthritis Associates of Southern Indiana, Jeffersonville, Indiana
  - Research Institute of Middle America/River Cities Cardiology, Jeffersonville, Indiana
  - Beacon Medical Group LaPorte, La Porte, Indiana
  - Cardiovascular Clinics, PC, Merrillville, Indiana
  - Community Clinical Research Center, Muncie, Indiana
  - Medical Specialists Clinical Research Center, Munster, Indiana
  - Medical Specialists, Munster, Indiana
  - Arthritis Associates of Southern Indiana, New Albany, Indiana
  - Buynak Clinical Research, Valparaiso, Indiana
  - Physician's Clinic of Iowa, PC, Cedar Rapids, Iowa
  - Ridge Family Practice, PC/Clinical Research Advantage, Inc., Council Bluffs, Iowa
  - Midwest Cardiovascular Research Foundation, Davenport, Iowa
  - Office of Jerrold V Flatt, Des Moines, Iowa
  - Medical Associates Clinic, PC, Dubuque, Iowa
  - Family Health Center of Waterloo, PC, Waterloo, Iowa
  - Northeast IA Medical Education Foundation/Family Practice Center, Waterloo, Iowa
  - Heartland Research Associates LLC, Arkansas City, Kansas
  - Community House of Wellness, Kansas City, Kansas
  - Associates Reseach Inc., Lansing, Kansas
  - Radiant Research, Inc., Overland Park, Kansas
  - International Clinical Research Institute, Inc, Overland Park, Kansas
  - Arthritis Specialists of Greater KC, Overland Park, Kansas
  - Pinnacle Medical Research, Overland Park, Kansas
  - Quivira Internal Medicine, Overland Park, Kansas
  - Health Science Research Center, Pratt, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Via Christi Clinic, Wichita, Kansas
  - Howard L. Feinberg, D.O., Ashland, Kentucky
  - Graves Gilbert Clinic, Bowling Green, Kentucky
  - Internal Medicine Research Association, Campbellsville, Kentucky
  - Center for Arthritis and Osteoporosis, Elizabethtown, Kentucky
  - Arthritis Center of Lexington, Lexington, Kentucky
  - Kentuckiana Center for Better Bone and Joint Health, Louisville, Kentucky
  - KY Research PLLC., Louisville, Kentucky
  - University Medical Associates, Louisville, Kentucky
  - Louisville Metabolic and Atherosclerosis Research Center, Louisville, Kentucky
  - Office of Gaurang B. Shah,MD, PSC, Richmond, Kentucky
  - Richmond Regional Research, Richmond, Kentucky
  - Chandler Family Practice, Bossier City, Louisiana
  - McFarland Family Clinic, Shreveport, Louisiana
  - TFD Research, LLC, Shreveport, Louisiana
  - Maine Research Associates, Auburn, Maine
  - Southern Maine Health Care, Biddeford, Maine
  - Central Maine Heart & Vascular Institute, Lewiston, Maine
  - Chesapeake CardioVascular Associates, Baltimore, Maryland
  - Midatlantic Cardiovascular Associates, Baltimore, Maryland
  - Midatlantic Cardiovascular Associates, PA, Baltimore, Maryland
  - Health Trends Research, LLC, Baltimore, Maryland
  - One Heart, LLC, Baltimore, Maryland
  - Midatlantic Cardiovascular Associates, Pa, Baltimore, Maryland
  - Saint Agnes HealthCare Incorporated, Baltimore, Maryland
  - Stephen R Smith, MD FACP, Baltimore, Maryland
  - MidAtlantic Cardiovascular Associates, PA, Baltimore, Maryland
  - Peter A. Holt, Baltimore, Maryland
  - Midatlantic Cardiovascular Associates PA, Bel Air, Maryland
  - Shah Associates MD, LLC, Charlotte Hall, Maryland
  - Cardiovascular Specialists, LLC, Columbia, Maryland
  - Johns Hopkins University, Columbia, Maryland
  - The Osteoporosis & Clinical Trials Center, Cumberland, Maryland
  - Arthritis Treatment Center, Frederick, Maryland
  - The Spine & Joint Center, Greenbelt, Maryland
  - Klein & Associates, MD, PA, Hagerstown, Maryland
  - Community Health Research, North East, Maryland
  - MD Medical Research, Oxon Hill, Maryland
  - Shah Associates, Prince Frederick, Maryland
  - Cardiac Associates, Shady Grove Adventist Hospital, Rockville, Maryland
  - The Center for Rheumatology and Bone Research, Rockville, Maryland
  - Rockville Internal Medicine Group, Rockville, Maryland
  - IRC Clinics, Towson, Maryland
  - Midatlantic Cardiovascular Associates, P.A., Westminster, Maryland
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Primary Care Cardiology Research, Ayer, Massachusetts
  - Genesis Clinical Research & Consulting, Fall River, Massachusetts
  - NECCR Internal Medicine and Cardiology Associates, LLC, Fall River, Massachusetts
  - Phase III Clinical Research, Fall River, Massachusetts
  - Pentucket Medical Associates, Incorporated, Haverhill, Massachusetts
  - Clinical Research Center of Cape Cod, Inc., Hyannis, Massachusetts
  - Charles River Medical Associates, Pchi, Natick, Massachusetts
  - Novex Clinical Research, LLC, New Bedford, Massachusetts
  - Northampton Internal Medicine Associates, PC, Northampton, Massachusetts
  - FutureCare Studies, Springfield, Massachusetts
  - Reliant Medical Group, Inc., Worcester, Massachusetts
  - Great Lakes Research Group, Incorporated, Bay City, Michigan
  - Professional Clinical Research-Benzonia, Benzonia, Michigan
  - Cadillac Clinical Research, Cadillac, Michigan
  - Livernois Family Medical Services, Detroit, Michigan
  - Office of Dr. Susan Courtnage, Eaton Rapids, Michigan
  - McLaren Regional Medical Center-Research Dept., Flint, Michigan
  - Grand Valley Medical Specialist, PLC, Grand Rapids, Michigan
  - Spectrum Health Medical Group-Rheumatology, Grand Rapids, Michigan
  - Michigan Medical Cardiovascular PC, Grand Rapids, Michigan
  - Professional Clinical Research, Interlochen, Michigan
  - Justus J Fiechtner, MD, Lansing, Michigan
  - Michigan Cardiovascular Institute, Saginaw, Michigan
  - Synergy Medical Education Alliance, Saginaw, Michigan
  - Shores Rheumatology, Saint Clair Shores, Michigan
  - Oakland Medical Research Center, Troy, Michigan
  - Troy Internal Medicine Research, Troy, Michigan
  - St. Luke's Hospital Association of Duluth, DBA St Luke's Rheumatology Assoc., Duluth, Minnesota
  - St. Luke's Hospital Association of Duluth, Inc., Duluth, Minnesota
  - St. Luke's Hospital Association of Duluth, Duluth, Minnesota
  - Central Minnesota Heart Center at St. Cloud Hospital, Saint Cloud, Minnesota
  - St. Paul Heart Clinic, Saint Paul, Minnesota
  - The Center for Clinical Trials, Biloxi, Mississippi
  - Planters Clinic, Port Gibson, Mississippi
  - North Mississippi Medical Clinics, Inc., Tupelo, Mississippi
  - Cape Girardeau Physicians Associates, Cape Girardeau, Missouri
  - Patterson Medical Clinic / d.b.a. Prime Care Research Associates, Florissant, Missouri
  - Allergy Asthma Immunology Services, LLC, Jefferson City, Missouri
  - Jefferson City Medical Group, Jefferson City, Missouri
  - University of Missouri Kansas City School of Medicine, Kansas City, Missouri
  - Truman Medical Center, Inc., Kansas City, Missouri
  - Clinical Research Advantage, Inc./Manning Family Care, LLC, Kansas City, Missouri
  - Mercy Medical Research Institute, Springfield, Missouri
  - St. Louis Center for Clinical Research, St Louis, Missouri
  - Physician Groups, LC, DBA Rheumatology and Internal Medicine Associates, St Louis, Missouri
  - Southampton Healthcare, Inc., St Louis, Missouri
  - Barbara A. Caciolo, MD, St Louis, Missouri
  - A & A Pain Institute, St Louis, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Patients First Health Care, LLC, Washington, Missouri
  - Glacier View Research Institute, Cardiology, Kalispell, Montana
  - Alliance Medical Center, Alliance, Nebraska
  - Cody Medical Associates, Alliance, Nebraska
  - Bellevue Family Practice/Clinical Research Advantage, Inc., Bellevue, Nebraska
  - Clinical Research Advantage, Inc./ Skyline Medical Center, PC, Elkhorn, Nebraska
  - Clinical Research Advantage, Inc./Prairie Fields Family Medicine, PC, Fremont, Nebraska
  - Internal Medicine Associates, PC, Grand Island, Nebraska
  - Physician, Research Collaboration, Southwest Family Health, Lincoln, Nebraska
  - Lincoln Internal Medicine Associates, Lincoln, Nebraska
  - Platte River Nephrology, North Platte, Nebraska
  - Quality Clinical Research LLC, Omaha, Nebraska
  - Westroads Medical Group, Omaha, Nebraska
  - Heartland Clinical Research, Inc., Omaha, Nebraska
  - Clinical Research Advantage, Inc./Primary Care Physicians, LLP, Omaha, Nebraska
  - Clinical Research Advantage, Inc., Henderson, Nevada
  - Clinical Research Advantage, Inc./Rita B. Chuang, MD, LLC, Henderson, Nevada
  - Sierra Internal Medicine Associates, Incline Village, Nevada
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - Clinical Research Advantage/Peter Philander, MD, Las Vegas, Nevada
  - Rancho Internal Medicine, Las Vegas, Nevada
  - Steven D. Folkerth, MD, Las Vegas, Nevada
  - Ladner Family Practice, Las Vegas, Nevada
  - VA Southern Nevada Healthcare System, North Las Vegas, Nevada
  - Arthritis Center of Reno, Reno, Nevada
  - New Jersey Physicians, LLC, Clifton, New Jersey
  - Clifton-Wallington Medical Group, Clifton, New Jersey
  - Anderson and Collins, Clinical Research Inc., Edison, New Jersey
  - Drs. Collins and Uthappa, Edison, New Jersey
  - Central Jersey Health Care, Elizabeth, New Jersey
  - Andron Medical Associates, Englewood, New Jersey
  - Advocare Heights Primary Care, Haddon Heights, New Jersey
  - Hazlet Health Care, Hazlet, New Jersey
  - Family Care Physicians, Lawrenceville, New Jersey
  - Penn Cardiac Care at Mercer Bucks, Lawrenceville, New Jersey
  - Family Medicine of Lindenwold, Lindenwold, New Jersey
  - Rheumatology and Arthritis Associates PC, Medford, New Jersey
  - Adult & Pediatric Rheumatology, Midland Park, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - Maynard Holgado LLC, Sicklerville, New Jersey
  - Shore Health Group, Toms River, New Jersey
  - Hopewell Valley Medical Group, P.A., Trenton, New Jersey
  - Arthritis, Rheumatic and Back Disease Associates, PA, Voorhees Township, New Jersey
  - Lourdes Medical Associates, Willingboro, New Jersey
  - Kenneth F. Solinsky, MD, Babylon, New York
  - LifeLine Research Institute, Brooklyn, New York
  - Lee Medical Associates, Dunkirk, New York
  - AMS Research, Elmira, New York
  - Regional Clinical Research, Inc., Endwell, New York
  - Drug Trials America, Inc., Hartsdale, New York
  - United Health Service Hospitals, Office of Clinical Trials, Johnson City, New York
  - IMA Medical Research PC, Kew Gardens, New York
  - NYU Langone Medical Center, Laura and Issac Perlmutter Cancer Center, Infusion Center, Lake Success, New York
  - NYU Langone Medical Center, Laura and Issac Perlmutter Cancer Center, Investigational Pharmacy, Lake Success, New York
  - NYU Langone Rheumatology Associates Long Island, Lake Success, New York
  - Office of Dr. Allen Chodock, Mamaroneck, New York
  - Winthrop University Hospital / Clinical Trials Center, Mineola, New York
  - New York University Pain Management Center, New York, New York
  - NYU Pain Research, New York, New York
  - Office of Dr. Richard Stern, New York, New York
  - DiGiovanna Family Care Center, North Massapequa, New York
  - Hudson Valley Heart Center, Poughkeepsie, New York
  - AAIR Research Center, Rochester, New York
  - Institute for Clinical Studies, Rosedale, New York
  - Rheumatology Associates of Long Island, Smithtown, New York
  - Office of Dr. Chadia Morcos, Syosset, New York
  - Arthritis Health Associates, Syracuse, New York
  - Crouse Medical Practice, PLLC d/b/a Internist Associates of Central New York, Syracuse, New York
  - East Meadow Family Practice Associates, PC, Wantagh, New York
  - Southgate Medical Group, West Seneca, New York
  - Great Lakes Medical Research, Westfield, New York
  - Buffalo Cardiology and Pulmonary Associates, PC, Williamsville, New York
  - Upstate Clinical Research Associates, Williamsville, New York
  - Asheville Arthritis & Osteoporosis, PA, Asheville, North Carolina
  - Kernodle Clinic Inc., Burlington, North Carolina
  - Calabash Medical Center, Calabash, North Carolina
  - PMG Research of Raleigh, LLC d/b/a PMG Research of Cary, Cary, North Carolina
  - Chapel Hill Family Medicine, Chapel Hill, North Carolina
  - Thurston Arthritis Reaserch Ctr, Chapel Hill, North Carolina
  - Mid Carolina Cardiology Research, Charlotte, North Carolina
  - Presbyterian Novant Heart and Wellness, Charlotte, North Carolina
  - Arthritis and Osteoporosis Consultants of the Carolinas, Charlotte, North Carolina
  - PMG Research of Charlotte, Charlotte, North Carolina
  - Barat Research Group, Inc., Charlotte, North Carolina
  - Sensenbrenner Primary Care, Charlotte, North Carolina
  - Duke Health Center at Pickett Road, Durham, North Carolina
  - Bland Clinic, PA, Greensboro, North Carolina
  - Medication Management, LLC, Greensboro, North Carolina
  - Physicians East P. A., Greenville, North Carolina
  - Physicians East, PA, Greenville, North Carolina
  - Clinical Trials of America, Inc., Hickory, North Carolina
  - PMG Research Of Hickory, LLC, Hickory, North Carolina
  - Peters Medical Research, High Point, North Carolina
  - Research Institute of the Carolinas, PLLC, Mooresville, North Carolina
  - Crystal Coast Family Practice, Morehead City, North Carolina
  - Burke Primary Care, Morganton, North Carolina
  - Pinehurst Medical Clinic, Inc., Pinehurst, North Carolina
  - Pinehurst Medical Clinic. Inc., Pinehurst, North Carolina
  - Blue Ridge Family Physicians, PPLC, Raleigh, North Carolina
  - PMG Research of Raleigh, LLC, Raleigh, North Carolina
  - Wake Internal Medicine Consultants, Inc., Raleigh, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Boice-Willis Clinic, Rocky Mount, North Carolina
  - PMG Research of Salisbury, Salisbury, North Carolina
  - Tabor City Family Medicine, Tabor City, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - PMG Research Wilmington Research Associates, Wilmington, North Carolina
  - Natalie A. Doyle, MD PA, Wilson, North Carolina
  - Ardmore Family Practice, Winston-Salem, North Carolina
  - Clinical Trials of America, Inc., Winston-Salem, North Carolina
  - Clinical Trials of America, inc, Winston-Salem, North Carolina
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
  - Winston-Salem Health Care, Winston-Salem, North Carolina
  - Plains Clinical Research Center, Fargo, North Dakota
  - Daystar Clinical Research, Akron, Ohio
  - CFP Research, Inc., Cincinnati, Ohio
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Feldman Family Practice, Columbus, Ohio
  - MidWest Cardiology Research Foundation, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Remington-Davis Incorporated, Columbus, Ohio
  - Midtowne Family Practice Centre, Columbus, Ohio
  - PriMed Clinical Research, Dayton, Ohio
  - HWC Women's Research Center, Englewood, Ohio
  - Cleveland Clinic Fairview Cardiovascular Medicine, Fairview Park, Ohio
  - Prestige Clinical Research, Franklin, Ohio
  - TriPhase Research, Ltd., Franklin, Ohio
  - Holzer Clinic, Inc, Gallipolis, Ohio
  - Office of Dr. Saleem Khan, MD, Inc, London, Ohio
  - North Central Research, Mansfield, Ohio
  - OhioHealth Research Institute, Mansfield, Ohio
  - R&R Research-Smith Clinic, Marion, Ohio
  - David R. Mandel, MD, Inc, Mayfield, Ohio
  - Paramount Medical Research and Consulting, LLC, Middleburg Heights, Ohio
  - Newark Physician Associates, Newark, Ohio
  - Family Medicine and Occupational Health Center, Inc., Shaker Heights, Ohio
  - Abner Cordero, M.D., Tiffin, Ohio
  - Arthritis Associates of Northwest Ohio, Inc., Toledo, Ohio
  - Mercy St Vincent Medical Center, Toledo, Ohio
  - Toledo Cardiology Consultants c/o Cardiac Research, Toledo, Ohio
  - South Toledo Internists, Toledo, Ohio
  - University of Toledo Health Science Campus, Toledo, Ohio
  - UT Medical Center Medicine Clinic, Toledo, Ohio
  - Trenton Family Medicine, Trenton, Ohio
  - Lake Medical Research, LLC, Willoughby Hills, Ohio
  - Pharmacotherapy Research Associates Incorporated, Zanesville, Ohio
  - LION Research, Norman, Oklahoma
  - Integris Physicians Services, Oklahoma City, Oklahoma
  - Integris Cardiovascular Physicians LLC, Oklahoma City, Oklahoma
  - Integris Family Care Central, Oklahoma City, Oklahoma
  - Integris Physician Services, Oklahoma City, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Healthcare Research Consultants, Tulsa, Oklahoma
  - Integrated Medical Research, PC, Ashland, Oregon
  - Lane Medical Research Group, Eugene, Oregon
  - Oregon Medical Group Adult Medicine Clinic, Eugene, Oregon
  - Oregon Medical Group Clinical Research, Eugene, Oregon
  - Institute of Diabetes and Endocrinology, Medford, Oregon
  - Rogue Valley Physicians-Clinical Research Group, Medford, Oregon
  - Fanno Creek Clinic, Portland, Oregon
  - Affinity Research, Portland, Oregon
  - Portland Rheumatology Clinic, LLC, Portland, Oregon
  - Internal Medicine Research, Portland, Oregon
  - University Orthopedics Center, Altoona, Pennsylvania
  - Tri-State Medical Group, Beaver, Pennsylvania
  - East Penn Rheumatology Associates, PC, Bethlehem, Pennsylvania
  - Buckingham Family Medicine, Buckingham, Pennsylvania
  - Camp Hill Clinical Research Center, Camp Hill, Pennsylvania
  - Butler Medical Associates, Chicora, Pennsylvania
  - Perkiomen Valley Family Practice, PC, Collegeville, Pennsylvania
  - Rheumatology Associates, Ltd, Colmar, Pennsylvania
  - Office of J. Miller Oppy, MD, Youghiogheny Primary Care Practice, Connellsville, Pennsylvania
  - Brandywine Clinical Research, Downingtown, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Saint Vincent Consultant in Cardiovascular Diseases, LLC, Erie, Pennsylvania
  - Arthritis Associates, Erie, Pennsylvania
  - Center for Assessment and Research of Erie, Erie, Pennsylvania
  - Stan F. Slabic, M.D., Erie, Pennsylvania
  - AMH Feasterville Family HealthCare Center, Feasterville, Pennsylvania
  - Westmoreland Neurology Associates, Incorporated, Greensburg, Pennsylvania
  - Harleysville Medical Assoc, Harleysville, Pennsylvania
  - Lederach Family Medicine, Harleysville, Pennsylvania
  - Dr. Bruce Morrison, Family Practice, Huntingdon Valley, Pennsylvania
  - Detweiler Family Medicine and Associates, PC, Lansdale, Pennsylvania
  - Green and Seidner Family Practice Associates, Lansdale, Pennsylvania
  - Lansdale Medical Group Family Practice, Lansdale, Pennsylvania
  - Bucks County Clinical Research, Morrisville, Pennsylvania
  - Pearl Clinical Research, Inc., Norristown, Pennsylvania
  - Lehigh Wellness Center Outpatient Services, Philadelphia, Pennsylvania
  - Founders Research Corporation, Philadelphia, Pennsylvania
  - VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - Dairyland Medical Center, Red Lion, Pennsylvania
  - Sfm Clinical Trials, PC, Scotland, Pennsylvania
  - Elite Medical Research, Inc., Sellersville, Pennsylvania
  - Prime Health Network, Springfield, Pennsylvania
  - University Orthopedics Center, State College, Pennsylvania
  - The Office of Dr. Joseph T. Morelli, DO, Stoneboro, Pennsylvania
  - Tipton Medical and Diagnostic Center, Tipton, Pennsylvania
  - Pish Medical Associates, Uniontown, Pennsylvania
  - PEAK Research, LLC, Upper Saint Clair, Pennsylvania
  - Allegheny Rheumatology - WPAHS - ASRI, Wexford, Pennsylvania
  - Clinical Research Center of Reading, LLC, Wyomissing, Pennsylvania
  - Cardiology Consultants of Philadelphia, Yardley, Pennsylvania
  - Jeffry A. Lindenbaum DO, PC, Yardley, Pennsylvania
  - New England Center for Clinical Research, Cranston, Rhode Island
  - Partners in Clinical Research, Cumberland, Rhode Island
  - Hugo M. Yamada, MD, Lincoln, Rhode Island
  - Rheumatology Associates, Pawtucket, Rhode Island
  - Medical Office Center, Providence, Rhode Island
  - Anderson Heart, Anderson, South Carolina
  - AnMed Health, Anderson, South Carolina
  - Low Country Rheumatology, PA/Low Country Research Center, Charleston, South Carolina
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - St. Andrews Medical, Charleston, South Carolina
  - Neem Research Group Inc., Columbia, South Carolina
  - Columbia Arthritis Center Pa, Columbia, South Carolina
  - MedTrial, Columbia, South Carolina
  - Clinical Research Associates, LLC, Florence, South Carolina
  - Palmetto Clinical Trial Services, LLC, Greenville, South Carolina
  - Paris View Family Practice, Greenville, South Carolina
  - John Milas, Greer, South Carolina
  - Radiant Research, Inc, Greer, South Carolina
  - DeGarmo Institute of Medical Research, Greer, South Carolina
  - Mountain View Clinical Research, Inc., Greer, South Carolina
  - Palmetto Clinical Trial Services, LLC at the Family Healthcare Center, Laurens, South Carolina
  - Berkeley Medical Center, Moncks Corner, South Carolina
  - PMG Research of Charleston, Mt. Pleasant, South Carolina
  - North Myrtle Beach Family Practice, North Myrtle Beach, South Carolina
  - Coulter Clinic, Orangeburg, South Carolina
  - Orangeburg Medical Associates, PA, Orangeburg, South Carolina
  - The Carolina Center for Rheumatology & Arthritis Care, PA, Rock Hill, South Carolina
  - Hillcrest Clinical Research, LLC, Simpsonville, South Carolina
  - Hillcrest Family Practice, Simpsonville, South Carolina
  - Palmetto Research, Spartanburg, South Carolina
  - Palmetto Clinical Research, Summerville, South Carolina
  - Southeastern Research Associates, Inc., Taylors, South Carolina
  - Odyssey Research/Sanford Clinic - Aberdeen, Aberdeen, South Dakota
  - Sanford Clinic - Aberdeen, Aberdeen, South Dakota
  - Regional Health Clinic Research, Rapid City, South Dakota
  - Regional Medical Clinic-Rheumatology, Rapid City, South Dakota
  - Health Concepts, Rapid City, South Dakota
  - Brown Clinic PLLP, Watertown, South Dakota
  - Odyssey Research, Watertown, South Dakota
  - Holston Medical Group, Bristol, Tennessee
  - Internal Medicine & Pediatric Associates of Bristol, Bristol, Tennessee
  - PMG Research of Bristol, Bristol, Tennessee
  - Parkway Medical Group, Fayetteville, Tennessee
  - Stern Cardiovascular Foundation, inc., Germantown, Tennessee
  - Arthritis Clinic, Jackson, Tennessee
  - The Jackson Clinic, PA, Jackson, Tennessee
  - State of Franklin Healthcare Associates Clinical Research, Johnson City, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Holston Valley Surgery Center, Kingsport, Tennessee
  - Gupta, Ramesh C MD, Memphis, Tennessee
  - Access Clinical Trials, Inc., Nashville, Tennessee
  - Premier Orthopaedics, Nashville, Tennessee
  - The Cholesterol Center of Nashville, Nashville, Tennessee
  - Nashville Medical Research Institute, Nashville, Tennessee
  - Quality Medical Research, Nashville, Tennessee
  - Amarillo Medical Specialists, LLP, Amarillo, Texas
  - Pharma Tex Research, LLC, Amarillo, Texas
  - Family Health Care Association, Arlington, Texas
  - South Arlington Primary Care Associates PA, Arlington, Texas
  - DCT - Anchor, LLC dba Discovery Clinical Trials, Arlington, Texas
  - DCT-AACT, LLC dba Discovery Clinical Trials, Austin, Texas
  - Southeast Texas Cardiology Associates, Beaumont, Texas
  - Southeast Texas Clinical Research Center, Beaumont, Texas
  - Kaner Medical Group PA, Bedford, Texas
  - Nexxus Research Group, LLC, Bedford, Texas
  - Texas Orthopedic Specialists, PLLC, Bedford, Texas
  - MedicalEdge Healthcare Group, PA, dba Leading Edge Research, PA, Carrollton, Texas
  - Prentiss Family Medicine, Colleyville, Texas
  - Carlos B. Everett, MD, Corpus Christi, Texas
  - Discovery Clinical Research, Corpus Christi, Texas
  - Texas Health Physicians Group, Dallas, Texas
  - Soltero Cardiovascular Research Center/Baylor University Medical Center, Dallas, Texas
  - Arthritis Care and Diagnostic Center, P.A., Dallas, Texas
  - Medical Specialists Associated, Dallas, Texas
  - Metroplex Clinical Research Center, Dallas, Texas
  - SouthWest Rheumatology, P.A., Dallas, Texas
  - DCT - Genesis Neighborhood Research, LLC dba Discovery Clinical Trials, Dallas, Texas
  - Rajendra K. Marwah, MD, El Paso, Texas
  - Kaner Medical Group, PA, Euless, Texas
  - The Medical Group of Texas, Fort Worth, Texas
  - Texas Health Physicians Group, Fort Worth, Texas
  - T & R Clinic, P. A., Fort Worth, Texas
  - Rheumatology-UTMB, Galveston, Texas
  - Towngate Plaza Medical Center, Garland, Texas
  - ProCare Clinical Trials, Grand Prairie, Texas
  - The Office of Amer Zaheer MD, PA, Houston, Texas
  - Salim Gopalani, MD, PA, Houston, Texas
  - Office of Cyril Wolf, MD, Houston, Texas
  - Village Family Practice, Houston, Texas
  - Kelsey Seybold Clinic, Houston, Texas
  - Oxford Clinical Research, LLC, Houston, Texas
  - MCA Research, Houston, Texas
  - Texas Health Physicians Group, Irving, Texas
  - One World Medical Associates, P.A., Lewisville, Texas
  - Pri-Med Care, Lewisville, Texas
  - South Texas Institute of Health, McAllen, Texas
  - DCT - Genesis Seidmeyer Research, LLC dba Discovery Clinical Trials, McKinney, Texas
  - Southwest Rheumatology, PA, Mesquite, Texas
  - Midland Clinical Research Center, Midland, Texas
  - Basin Orthopedics Surgical Specialists, Odessa, Texas
  - Center for Hypertension and Internal Medicine, Odessa, Texas
  - Odessa Heart Institute, Odessa, Texas
  - Permian Research Foundation, Odessa, Texas
  - Office of David K. McDonald, M.D.. P.A., Pasadena, Texas
  - Centex Studies, Inc., Pharr, Texas
  - Clinical Investigations of Texas, LLC, Plano, Texas
  - DCT-Genesis naini, LLC dba Discovery Clinical Trials, Plano, Texas
  - North Texas Medical Research, Plano, Texas
  - MedicalEdge Healthcare Group, PA, Richardson, Texas
  - Texas Health Physicians Group, Richardson, Texas
  - Ivan N. Mefford, MD, PhD, PA, Richmond, Texas
  - Paragon Research Center, LLC, San Antonio, Texas
  - Quality Assurance Research Center, San Antonio, Texas
  - Quality Research Inc., San Antonio, Texas
  - Physician PrimeCare Research Institute, PLLC dba Health Texas Research Institute, San Antonio, Texas
  - GSA Research, San Antonio, Texas
  - Sun Research Institute, San Antonio, Texas
  - Radiant Research San Antonio Northeast, San Antonio, Texas
  - Briggs Clinical Research, LLC, San Antonio, Texas
  - DCT - Barlite, LLC dba Discovery Clinical Trials, San Antonio, Texas
  - S.A.M. Clinical Research Center, San Antonio, Texas
  - WellMed Clinical Research, San Antonio, Texas
  - DCT-Westover Hills, LLC dba Discovery Clinical Trials, San Antonio, Texas
  - DCT - Stone Oak, LLC dba Discovery Clinical Trials, San Antonio, Texas
  - The Office of Shahbaz Yazdani, MD, PA, San Antonio, Texas
  - Southlake Clinical Trials, Southlake, Texas
  - Sugar Land Med-Ped Clinic, PA, Sugar Land, Texas
  - Crossroads Clinical Research, LLC, Victoria, Texas
  - Crossroads Clinical Research, Victoria, Texas
  - Office of Pamela Dugano-Daphnis, Webster, Texas
  - Advanced Research Institute, Ogden, Utah
  - Advanced Clinical Research, West Jordan, Utah
  - Burke Internal Medicine & Research, Burke, Virginia
  - Burke Internal Medicine, Burke, Virginia
  - Center for Arthritis and Rheumatic Diseases, Chesapeake, Virginia
  - Bayview Physicians oa Cardiovascular Associates, Ltd, Chesapeake, Virginia
  - David Ramstad, MD, MPH and Associates, Chesapeake, Virginia
  - Danville Internal Medicine, Inc., Danville, Virginia
  - Danville Orthopedic Clinic, Danville, Virginia
  - Seven Corners Medical Research Center, Falls Church, Virginia
  - Hampton Family Practice, Hampton, Virginia
  - Manassas Clinical Research Center, Manassas, Virginia
  - Bruton Avenue Family Practice, Newport News, Virginia
  - Internal Medicine Kidney and Hypertension Center, Norfolk, Virginia
  - National Clinical Research - Norfolk Inc., Norfolk, Virginia
  - Sentara Medical Group, Norfolk, Virginia
  - Ettrick Health Center, Petersburg, Virginia
  - Arthritis and Rheumatic Research, Portsmouth, Virginia
  - Roanoke Heart Institute, Roanoke, Virginia
  - Harbourview Professional Center, Suffolk, Virginia
  - Chase Research Group, LLC, Virginia Beach, Virginia
  - The Center for Excellence in Aging and Geriatric Health, Williamsburg, Virginia
  - Highline Medical Center Laboratory, Burien, Washington
  - Puget Sound Osteoporosis Center, Seattle, Washington
  - Arthritis Northwest, Seattle, Washington
  - Arthritis Northwest Rheumatology, Spokane, Washington
  - Lawrence S. Eastburn, MD, PS, Spokane, Washington
  - Pulmonary and Research Associates, Spokane, Washington
  - The Office of William Gray, Md, Family Practice, Spokane, Washington
  - John F. Long, D.O., Spokane, Washington
  - George H. Krick, MD, Tacoma, Washington
  - Northwest Family and Spinal Clinic, Tacoma, Washington
  - Rheumatology Infusion Services, Tacoma, Washington
  - Tacoma Center for Arthritis Research, PS, Tacoma, Washington
  - Wenatchee Valley Medical Center, Research Department, Wenatchee, Washington
  - Clinical Trials Northwest, Yakima, Washington
  - Rheumatology and Pulmonary Clinic, Beckley, West Virginia
  - Mountain State Clinical Research, Clarksburg, West Virginia
  - University Cardiovascular Services. Robert C. Byrd Clinical Center, Huntington, West Virginia
  - WVVA Healthcare Alliance, Lewisburg, West Virginia
  - Parkersburg Cardiology Associates, Parkersburg, West Virginia
  - Meriter Medical Group, Madison, Wisconsin
  - University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin
  - UW Health Physicians, Madison, Wisconsin
  - St. Lukes Pain Management Center, Milwaukee, Wisconsin
  - Zablocki VA Medical Center, Milwaukee, Wisconsin
  - Aspirus Cardiovascular Associates - Rhinelander, Rhinelander, Wisconsin
  - Aspirus Cardiovascular Associates, Wausau, Wisconsin
  - Aspirus Heart & Vascular lnstitute--Research & Education), Wausau, Wisconsin
  - Aspirus Wausau Hospital, Wausau, Wisconsin
  - Allegiance Research Specialists, LLC, Wauwatosa, Wisconsin
- Australia (12):
  - Hunter Clinical Research, Broadmeadow, New South Wales
  - Wesley Medical Centre, Auchenflower, Queensland
  - Australian Clinical Research Organisation, Caboolture, Queensland
  - Rheumatology Department, Cairns, Queensland
  - AusTrials Pty Ltd, Kippa-Ring, Queensland
  - Core Research Group, Milton, Queensland
  - AusTrials Pty Ltd, Sherwood, Queensland
  - Monash Medical Centre, Department of Rheumatology, Clayton, Victoria
  - Rheumatology Department, Heidelberg West, Victoria
  - Emeritus Research, Malvern East, Victoria
  - The Goatcher Clinical Research Unit, Shenton Park, Western Australia
  - The Colin Bayliss Research and Teaching Unit, Victoria Park, Western Australia
- Brazil (33):
  - CLINCOR - Clinica de Exames Cardiologicos e Ecografia S/C Ltda, Maceió, Alagoas
  - Hospital do Coracao de Alagoas, Maceió, Alagoas
  - CIP - Centro Internacional de Pesquisas, Goiânia, Goiás
  - Via Medica - Centro Clinico, Goiânia, Goiás
  - Hopsital das Clinicas da Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais
  - CMIP - Centro Mineiro de Pesquisa, Juiz de Fora, Minas Gerais
  - Hospital e Maternidade Angelina Caron, Sala Pesquisa Clinica, Campina Grande do Sul, Paraná
  - CEPEME-CERHFAC Centro de Estudos e Pesquisas Medicas, Curitiba, Paraná
  - Centro de Estudos do Hospital de Clínicas da UFPR, Curitiba, Paraná
  - Hospital Universitário Clementino Fraga Filho - UFRJ, Rio de Janeiro, Rio de Janeiro
  - CCBR Brasil Centro de Pesquisas e Analises Clinicas Ltda, Rio de Janeiro, Rio de Janeiro
  - Hospital Ipanema Plus, Rio de Janeiro, Rio de Janeiro
  - Clinica de Reumatologia do Centro Médico BarraShopping, Rio de Janeiro, Rio de Janeiro
  - Centro de Pesquisa Clinica, Porto Alegre, Rio Grande do Sul
  - Associação Hospitalar Moinhos de Vento (AHMV) / CMIC, Porto Alegre, Rio Grande do Sul
  - Hospital São Lucas - Pontificia, Porto Alegre, Rio Grande do Sul
  - Centro de Ensino e Pesquisa Hospital Sao Lucas, Aracaju, Sergipe
  - Hospital e Maternidade Celso Pierro - Puc Campinas, Campinas, São Paulo
  - PUC Campinas, Campinas, São Paulo
  - Hospital das Clinicas da UNICAMP, Campinas, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina de Marilia, Marília, São Paulo
  - Hospital de Base - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - CPCLIN - Centro de Pesquisas Clínicas, São Paulo, São Paulo
  - Hospital Alemao Oswaldo Cruz, São Paulo, São Paulo
  - Setor de Lip., Arterosc. e BioVasc. - Disc. de Cardiologia, São Paulo, São Paulo
  - CEPIC - Centro Paulista de Investigacao Clínica, São Paulo, São Paulo
  - IMA Brasil - Instituto de Medicina Avancada, São Paulo, São Paulo
  - Hospital Sao Salvador - Medicos Reunidos Ltda., Goiania-GO
  - Ambulatorio de Especialidades Mario Covas, Marilia/SP
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, RS
  - Hospital das Clinicas da UFPE, Recife - Pernambuco
  - Hospital Dos Servidores Do Estado do Rio de Janeiro, Rio de Janeiro
  - Faculdade de Medicina DO ABC, Santo André
- Canada (67):
  - South Calgary Medical Clinic - Sunpark Professional Center, Calgary, Alberta
  - Allin Clinic, Edmonton, Alberta
  - Dr. MPJ Senaratne Professional Corporation, Edmonton, Alberta
  - Medical Arts Health Research Group, Kelowna, British Columbia
  - The Medical Arts Health Research Group, Penticton, British Columbia
  - Ocean West Research Clinic Inc., Surrey, British Columbia
  - Prohealth Clinical Research Inc., Vancouver, British Columbia
  - Office of Dr. Milton F. Baker, Victoria, British Columbia
  - The Medical Arts Health Research Group, West Vancouver, British Columbia
  - Rivergrove Medical Clinic, Winnipeg, Manitoba
  - Manitoba Clinic, Winnipeg, Manitoba
  - G.A. Research Associates Ltd/Ltee, Moncton, New Brunswick
  - Eric N. Grant Professional Corporation, Quispamis, New Brunswick
  - Office of Dr. Brian N. Craig, Saint John, New Brunswick
  - Commonwealth Medical Clinic, Mount Pearl, Newfoundland and Labrador
  - Paradise Medical Clinic, Paradise, Newfoundland and Labrador
  - White Hills Medical Clinic, St. John's, Newfoundland and Labrador
  - Nexus Clinic Research, St. John's, Newfoundland and Labrador
  - The Clinical Trials Centre, St. John's, Newfoundland and Labrador
  - Topsail Road Medical Clinic, St. John's, Newfoundland and Labrador
  - MSHJ Research Associates, Inc., Halifax, Nova Scotia
  - Colchester Research Group, Truro, Nova Scotia
  - Office of Dr. Rohit Nagpal, Brampton, Ontario
  - Aggarwal and Associates Ltd., Brampton, Ontario
  - Aviva Clinical Trial Group Inc., Burlington, Ontario
  - Corunna Medical Research Center, Corunna, Ontario
  - C & L Research, Fort Erie, Ontario
  - Office of Dr. Swaran K. Syan, Greater Sudbury, Ontario
  - Office of Dr. Jonathan D. Adachi, Hamilton, Ontario
  - Office of Dr. John Mutrie, Kitchener, Ontario
  - KW Musculoskeletal Research Inc., Kitchener, Ontario
  - East London Medical Centre, London, Ontario
  - London East Medical Centre, London, Ontario
  - Office of Dr. Gordon Schacter, London, Ontario
  - Office of Dr. William Blake Bowler, London, Ontario
  - Office of Dr. Robert G. Luton, London, Ontario
  - Malton Medical Centre, Mississauga, Ontario
  - The Arthritis Program Research Group Inc., Newmarket, Ontario
  - SKDS Research Inc., Newmarket, Ontario
  - Office of Dr. Azim M. Velji, Niagara Falls, Ontario
  - AIM Health Group Trainyards Health and Wellness Centre, Ottawa, Ontario
  - London Road Diagnostic Clinic & Medical Center, Sarnia, Ontario
  - London Road Diagnostic Clinic & Medical Centre, Sarnia, Ontario
  - Keele Medical Place, Toronto, Ontario
  - Prime Health Clinical Research, Toronto, Ontario
  - Office of Dr. Ira Bernstein, Toronto, Ontario
  - Office of Dr. Subodh Kanani, Toronto, Ontario
  - Manna Research, Toronto, Ontario
  - North Walkerville Orthopaedic Associates, Windsor, Ontario
  - Research Office, Windsor, Ontario
  - Clinical Research and Arthritis Centre, Windsor, Ontario
  - Centre de sante et de services sociaux de Chicoutimi, Chicoutimi, Quebec
  - ECOGENE-21 / Centre de sante et de services sociaux de Chicoutimi, Chicoutimi, Quebec
  - Clinique de Medicine Familiale de Cowansville, Cowansville, Quebec
  - Centre de recherche clinique Adapra Inc., L'Ancienne-Lorette, Quebec
  - Centre de Recherche Hochelaga/ Clinique Medicale Hochelaga, Montreal, Quebec
  - Recherche Medicale Appliquee Informatics (AMIR) Inc., Montreal, Quebec
  - Kells Medical Research Group, Inc., Pointe-Claire, Quebec
  - Recherche Clinique Sigma, Inc., Québec, Quebec
  - Le Manoir de l'Atrium, Québec, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec, Quebec
  - Clinique Services Sante Rosemere, Rosemère, Quebec
  - St-Jerome Medical Research Inc., Saint-Jérôme, Quebec
  - Centre Medical des Carrieres, Saint-Marc-des-Carrieres, Quebec
  - Centre de Recherche Musculo-Squelettique, Trois-Rivières, Quebec
  - Cardiology and Research, Westmount, Quebec
  - Downtown Medical Specialists, Saskatoon, Saskatchewan
- Colombia (7):
  - Hospital Pablo Tobon Uribe - Unidad de Investigaciones, Medellín, Antioquia
  - Reumalab S.A.S., Medellín, Antioquia
  - IPS Rodrigo Botero S.A.S., Medellín, Antioquia
  - Fundacion Cardioinfantil, Bogota, Cundinamarca
  - Clinica Colsanitas Sa, Bogota, Cundinamarca
  - Fundacion Cardiovascular de Colombia, Floridablanca, Santander Department
  - Fundacion Valle del Lili, Cali
- Costa Rica (16):
  - Clínica Vía San Juan, La Union de Tres Rios, Cartago Province
  - Clinica San Agustin, Desamparados Centro, Provincia de San José
  - Hospital CIMA San Jose, Escazú, Provincia de San José
  - Hospital Hotel La Catolica, Guadalupe, Provincia de San José
  - Consultorio Privado Dr. Alberto Lainez Ventosilla, Moravia, Provincia de San José
  - Centro Medico San Rafael, Alajuela
  - Centro de Reumatologia y Osteoporosis, Cartago
  - Clínica Garzona, Cartago
  - Clinica de Especialidades Medicas Drs. Saenz Castro, Heredia
  - Clínica Monte Sión, Heredia
  - Clínica San Antonio, Heredia
  - Centro Medico San Jose, San José
  - Edificio Panda, San José
  - Hospital Clinica Biblica, San José
  - Hospital Clínica Biblica, San José
  - Oficina Privada, San José
- Hong Kong (4):
  - Prince of Wales Hospital, Shatin, NEW Territories
  - Centre for Assessment and Treatment of Rheumatic Diseases, Department of Medicine and Geriatrics, New Territories, NT
  - Department of Medicine, Queen Mary Hospital, Pokfulam
  - Department of Medicine, North District Hospital, Sheung Shui, NT
- Mexico (11):
  - Comite Mexicano para la Prevencion de la Osteoporosis, A.C., México, D.F.
  - Instituto Mexicano de Investigación Clínica, S.A. de C.V, México, D.F.
  - Centro de Investigacion del Noroeste SC, Tijuana, Estado de Baja California
  - Hospital Regional ISSSTE, León, Guanajuato
  - Instituto Jalisciense de Investigación Clínica SA de CV, Guadalajara, Jalisco
  - Centro de Estudios de Investigacion Basica y Clinica SC., Guadalajara, Jalisco
  - CIF-BIOTEC, Medica Sur, Mexico City, Mexico City
  - Unidad de Investigacion Dr. Mario Alvizouri Muñoz Ac Del Hospital General Dr. Miguel Silva, Morelia, Michoacán
  - Hospital Central "Dr. Ignacio Morones Prieto" Unidad Regional de Reumatologia y Osteoporosis, San Luis Potosí City, San Luis Potosí
  - Centro Medico Toluca, Metepec, State of Mexico
  - Clinicos Asociados BOCM, S.C., Mexico City
- Centro de Investigación Marbella, Panama City, Panama
- Peru (6):
  - IPC - Centro de Salud Integral S.A., San Isidro, Lima region
  - Centro Empresarial - Altavista Polo 4, Santiago de Surco, Lima region
  - Instituto de Ginecologia y Reproducción & Cirugia Minimamente Invasiva, Santiago de Surco, Lima region
  - Clinica San Felipe, Lima
  - Centro de Investigaciones Medical, Lima
  - Clinica San Juan Bautista, Lima
- Philippines (8):
  - Mary Mediatrix Medical Center, Lipa City, Batangas
  - De La Salle Health Sciences Institute, Dasmariñas, Cavite
  - Chong Hua Hospital, Cebu City
  - Southern Philippines Medical Center, Davao City
  - Jose R. Reyes Memorial Medical Center, Manila
  - Chinese General Hospital and Medical Center, Manila
  - Hospital Research Unit, University of Santo Tomas Hospital, Manila
  - St. Luke's Medical Center, Quezon City
- Taiwan (11):
  - Chang Gung Memorial Hospital-Kaohsiung branch, Section of Allergy, Immunology, Nio Sung Township, Kaohsiung County
  - Tri-Service General Hospital, Neihu District, Taipei CITY
  - Buddhist Tzu Chi Dailin General Hospital, Chia-Yi County, Taiwan
  - Chang Gung Medical Foundation-Linkou Branch, Gueishan Township, Taoyuan County
  - Chi-Mei Medical Center, Tainan, YUNG KANG
  - Chung-Ho Memorial Hospital, Kaoshiung Medical University Hospital, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Tri-service General Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Ukraine (19):
  - CRI "Clinical Territorial Medical Association "University Clinic",, Simferopol, Autonomous Republic of Crimea
  - Municipal Medical Institution "City Clinical Hospital #3", Department of Rheumatology, Chernivtsi
  - MI Dnipropetrovsk Regional Clinical Hospital named after I.I Mechnikov, Dnipropetrovsk
  - State Institution "Dnipropetrovsk Medical Academy of MOH, Ukraine, Dnipropetrovsk
  - Rheumatology Department, MMI "City Clinical Hospital #5", DNMU n.a. M.Gorkyy,, Donetsk
  - Donetsk National Med University, Chair of Propaedeutics and Internal Medicine, Donetsk
  - Municipal Establishment of Health Care, Kharkiv
  - City Clinical Hospital # 8, Dept of Cardiology and Functional Diagnostics, Kharkiv
  - City Clinical Hospital #1, Kyiv
  - National Scientific Center "The Strazhesko Institute of Cardiology", Kyiv
  - State Institution "Republican clinical hospital of MOH of Ukraine", Kyiv
  - Family Medicine Department of NMAPE named after PL Shupyk,, Kyiv
  - Lutsk City Clinical Hospital, Lutsk
  - Municipal City Clinical Hospital #5, Lviv
  - Center of Reconstructive and Regenerative Medicine (University clinic) of, Odesa
  - Treatment-and-Diagnostic Center LLC "Desna" Ltd, Ternopil
  - Municipal enterprise " City Hospital # 7",, Zaporizhzhia
  - Municipal Institution "Zaporizhzhya City Multiple Discipline Clinical Hospital #9", Zaporizhzhya
  - Zhytomyr Regional Clinical Hospital n.a. O.F. Gerbachevs'kyy/ Rheumatology Center, Zhytomyr

REFERENCES:
- [Derived] Obeid S, Libby P, Husni E, Wang Q, Wisniewski LM, Davey DA, Wolski KE, Xia F, Bao W, Walker C, Ruschitzka F, Nissen SE, Luscher TF. Cardiorenal risk of celecoxib compared with naproxen or ibuprofen in arthritis patients: insights from the PRECISION trial. Eur Heart J Cardiovasc Pharmacother. 2022 Sep 3;8(6):611-621. doi: 10.1093/ehjcvp/pvac015. PMID 35234840
- [Derived] Chirikov VV, Walker C, Stephens JM, Schepman P, Chambers R, Bakir M, Poorman GW, Haider S, Farghaly M. Evaluating the Cost-Effectiveness of Celecoxib versus Ibuprofen and Naproxen in Patients with Osteoarthritis in United Arab Emirates Based on the PRECISION Trial. Clinicoecon Outcomes Res. 2021 May 19;13:409-420. doi: 10.2147/CEOR.S280556. eCollection 2021. PMID 34040400
- [Derived] Bao W, Gaffney M, Pressler ML, Fayyad R, Wisemandle W, Beckerman B, Wolski KE, Nissen SE. Strengthening the interpretability of clinical trial results by assessing the effect of informative censoring on the primary estimand in PRECISION. Clin Trials. 2020 Oct;17(5):535-544. doi: 10.1177/1740774520934747. Epub 2020 Jul 9. PMID 32643966
- [Derived] Solomon DH, Shao M, Wolski K, Nissen S, Husni ME, Paynter N. Derivation and Validation of a Major Toxicity Risk Score Among Nonsteroidal Antiinflammatory Drug Users Based on Data From a Randomized Controlled Trial. Arthritis Rheumatol. 2019 Aug;71(8):1225-1231. doi: 10.1002/art.40870. Epub 2019 Jun 12. PMID 30801994
- [Derived] Reed GW, Abdallah MS, Shao M, Wolski K, Wisniewski L, Yeomans N, Luscher TF, Borer JS, Graham DY, Husni ME, Solomon DH, Libby P, Menon V, Lincoff AM, Nissen SE. Effect of Aspirin Coadministration on the Safety of Celecoxib, Naproxen, or Ibuprofen. J Am Coll Cardiol. 2018 Apr 24;71(16):1741-1751. doi: 10.1016/j.jacc.2018.02.036. PMID 29673465
- [Derived] Solomon DH, Husni ME, Wolski KE, Wisniewski LM, Borer JS, Graham DY, Libby P, Lincoff AM, Luscher TF, Menon V, Yeomans ND, Wang Q, Bao W, Berger MF, Nissen SE; PRECISION Trial Investigators. Differences in Safety of Nonsteroidal Antiinflammatory Drugs in Patients With Osteoarthritis and Patients With Rheumatoid Arthritis: A Randomized Clinical Trial. Arthritis Rheumatol. 2018 Apr;70(4):537-546. doi: 10.1002/art.40400. PMID 29266879
- [Derived] Ruschitzka F, Borer JS, Krum H, Flammer AJ, Yeomans ND, Libby P, Luscher TF, Solomon DH, Husni ME, Graham DY, Davey DA, Wisniewski LM, Menon V, Fayyad R, Beckerman B, Iorga D, Lincoff AM, Nissen SE. Differential blood pressure effects of ibuprofen, naproxen, and celecoxib in patients with arthritis: the PRECISION-ABPM (Prospective Randomized Evaluation of Celecoxib Integrated Safety Versus Ibuprofen or Naproxen Ambulatory Blood Pressure Measurement) Trial. Eur Heart J. 2017 Nov 21;38(44):3282-3292. doi: 10.1093/eurheartj/ehx508. PMID 29020251
- [Derived] Nissen SE, Yeomans ND, Solomon DH, Luscher TF, Libby P, Husni ME, Graham DY, Borer JS, Wisniewski LM, Wolski KE, Wang Q, Menon V, Ruschitzka F, Gaffney M, Beckerman B, Berger MF, Bao W, Lincoff AM; PRECISION Trial Investigators. Cardiovascular Safety of Celecoxib, Naproxen, or Ibuprofen for Arthritis. N Engl J Med. 2016 Dec 29;375(26):2519-29. doi: 10.1056/NEJMoa1611593. Epub 2016 Nov 13. PMID 27959716

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 950 centers in Australia (11), Brazil (30), Canada (64), Colombia (7), Costa Rica (12), Hong Kong (4), Mexico (11), Panama (2), Peru (5), Philippines (8), Taiwan (10), Ukraine 19), and United States (767); a total of 24 sites were activated but did not randomized any subject.
Pre-assignment Details: All eligible participants were enrolled in to the study.
Groups:
- Celecoxib: Celecoxib 100-200 mg twice daily with placebo to match ibuprofen 600-800 mg thrice daily and placebo to match naproxen 375-500 mg twice daily
- Ibuprofen: Ibuprofen 600-800 mg thrice daily with placebo to match celecoxib 100-200 mg twice daily and placebo to match naproxen 375-500 mg twice daily
- Naproxen: Naproxen 375-500 mg twice daily with placebo to match celecoxib 100-200 mg twice daily and placebo to match ibuprofen 600-800 mg thrice daily.
Period: Overall Study
Arm/Group | Celecoxib | Ibuprofen | Naproxen
Started | 8072 | 8040 | 7969
Completed | 5664 | 5580 | 5621
Not Completed | 2408 | 2460 | 2348
Not completed — Other | 181 | 231 | 205
Not completed — No longer willing to participate | 600 | 606 | 585
Not completed — Withdrawal by Subject | 661 | 692 | 651
Not completed — Lost to Follow-up | 611 | 588 | 542
Not completed — Physician Decision | 80 | 76 | 59
Not completed — Does not meet entrance criteria | 13 | 10 | 8
Not completed — Death | 189 | 192 | 228
Not completed — Study terminated by sponsor | 11 | 4 | 8
Not completed — Missing Subject Summary Status | 62 | 61 | 62

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Celecoxib | Ibuprofen | Naproxen | Total
Number analyzed (Participants) | 8072 | 8040 | 7969 | 24081
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.0 (9.5) | 63.2 (9.4) | 63.3 (9.4) | 63.2 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5175 | 5174 | 5096 | 15445
  Male | 2897 | 2866 | 2873 | 8636

OUTCOME MEASURES:

1. Primary Outcome: The First Occurrence of Antiplatelet Trialists Collaboration (APTC) Composite Endpoint, Confirmed by the Clinical Events Committee (CEC).
Description: APTC events are defined as a composite of any of the following events: Death due to CV causes (including cardiac, cerebrovascular, venous thromboembolic, haemorrhagic, other vascular, or unknown cause); Non-fatal MI; Non-fatal stroke (including intracranial hemorrhages, stroke of ischemic or unknown etiology).
Time Frame: Intent to Treat (ITT) Population - 30 months; Modified ITT (MITT) Population - 42 months
Population: ITT - The ITT population will consist of all subjects randomized for participation in the study.
  MITT - The MITT analysis population consisted of all randomized subjects who had received at least one dose of study drug, and contributed at least one post-baseline visit.
Measure: Number; unit: Percentage of Partcipants
Arm/Group | Celecoxib | Ibuprofen | Naproxen
Number analyzed (Participants) | 8072 | 8040 | 7969
Percentage of Partcipants
  ITT (N = 8072, 8040, 7969) | 2.3 | 2.7 | 2.5
  MITT (N = 8030, 7990, 7933) | 1.7 | 1.9 | 1.8
Statistical Analysis 1: Comparison: Celecoxib vs Naproxen; ITT Population; Test type: Non-Inferiority or Equivalence — Non inferiority required a hazard ratio of 1.12 or lower, as well as an upper 95% confidence limit of 1.33 or lower in the ITT population and of 1.40 or lower in the MITT population; p = 0.0002, Regression, Cox — Non inferiority P value, α=0.025; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.76 to 1.13]
Statistical Analysis 2: Comparison: Celecoxib vs Naproxen; MITT Population; Test type: Non-Inferiority or Equivalence — Non-inferiority requires the hazard ratio does not exceed 1.12, and the upper bound of the two-sided 95% CI for the hazard ratio estimate does not exceed 1.40; p = 0.0001, Regression, Cox — Non inferiority P value, α=0.025; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.72 to 1.14]
Statistical Analysis 3: Comparison: Celecoxib vs Ibuprofen; ITT Population; Test type: Non-Inferiority or Equivalence — Non-inferiority requires the hazard ratio does not exceed 1.12, and the upper bound of the two-sided 95% CI for the hazard ratio estimate does not exceed 1.33; p < 0.0001, Regression, Cox — Non inferiority P value, α=0.025; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.70 to 1.04]
Statistical Analysis 4: Comparison: Celecoxib vs Ibuprofen; MITT Population; Test type: Non-Inferiority or Equivalence — Non-inferiority requires the hazard ratio does not exceed 1.12, and the upper bound of the two-sided 95% CI for the hazard ratio (HR) estimate does not exceed 1.40; p < 0.0001, Regression, Cox — Non-inferiority P-value, α=0.025; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.64 to 1.02]
Statistical Analysis 5: Comparison: Ibuprofen vs Naproxen; ITT Population; Test type: Non-Inferiority or Equivalence — Non-inferiority requires the hazard ratio does not exceed 1.12, and the upper bound of the two-sided 95% CI for the hazard ratio (HR) estimate does not exceed 1.33; p = 0.0182, Regression, Cox — Non-inferiority P-value, α=0.025; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.89 to 1.31]
Statistical Analysis 6: Comparison: Ibuprofen vs Naproxen; MITT Population; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 4]; p = 0.0250, Regression, Cox — Non-inferiority P-value, α=0.025; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.89 to 1.40]

2. Secondary Outcome: The First Occurrence of a Major Adverse Cardiovascular Events (MACE)
Description: MACE defined as the composite of CV death (including hemorrhagic death), non-fatal MI, non-fatal stroke, hospitalization for UA, revascularization or hospitalization for TIA
Time Frame: ITT Population - 30 months; MITT Population - 42 months
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Celecoxib | Ibuprofen | Naproxen
Number analyzed (Participants) | 8072 | 8040 | 7969
Percentage of Participants
  ITT (N = 8072, 8040, 7969) | 4.2 | 4.8 | 4.3
  MITT (N = 8030, 7990, 7933) | 3.1 | 3.6 | 3.2
Statistical Analysis 1: Comparison: Celecoxib vs Naproxen; ITT Population; Test type: Superiority or Other; p = 0.6427, Regression, Cox; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.83 to 1.12]
Statistical Analysis 2: Comparison: Celecoxib vs Ibuprofen; ITT Population; Test type: Superiority or Other; p = 0.0597, Regression, Cox; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.75 to 1.01]
Statistical Analysis 3: Comparison: Ibuprofen vs Naproxen; ITT Population; Test type: Superiority or Other; p = 0.1481, Regression, Cox; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.96 to 1.29]
Statistical Analysis 4: Comparison: Celecoxib vs Naproxen; MITT Population; Test type: Superiority or Other; p = 0.5758, Regression, Cox; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.80 to 1.13]
Statistical Analysis 5: Comparison: Celecoxib vs Ibuprofen; MITT Population; Test type: Superiority or Other; p = 0.0204, Regression, Cox; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.69 to 0.97]
Statistical Analysis 6: Comparison: Ibuprofen vs Naproxen; MITT Population; Test type: Superiority or Other; p = 0.0751, Regression, Cox; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.98 to 1.38]

3. Secondary Outcome: The First Occurrence of Clinically Significant Gastrointestinal Events (CSGIE)
Description: CSGIE include: Gastroduodenal (GD) hemorrhage, Gastric outlet obstruction, Gastroduodenal, small bowel or large bowel perforation, Large bowel hemorrhage, Small bowel hemorrhage, Acute GI hemorrhage of unknown origin, including presumed small bowel hemorrhage, Symptomatic gastric or duodenal ulcer
Time Frame: ITT Population - 30 months; MITT Population - 42 months
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Celecoxib | Ibuprofen | Naproxen
Number analyzed (Participants) | 8072 | 8040 | 7969
Percentage of Participants
  ITT (N = 8072, 8040, 7969) | 0.7 | 0.9 | 0.7
  MITT (N = 8030, 7990, 7933) | 0.3 | 0.7 | 0.7
Statistical Analysis 1: Comparison: Celecoxib vs Naproxen; ITT Population; Test type: Superiority or Other; p = 0.8576, Regression, Cox; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.67 to 1.40]
Statistical Analysis 2: Comparison: Celecoxib vs Ibuprofen; ITT Population; Test type: Superiority or Other; p = 0.1202, Regression, Cox; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.53 to 1.08]
Statistical Analysis 3: Comparison: Ibuprofen vs Naproxen; ITT Population; Test type: Superiority or Other; p = 0.1734, Regression, Cox; Hazard Ratio (HR) = 1.27, 95% CI 2-sided [0.90 to 1.81]
Statistical Analysis 4: Comparison: Celecoxib vs Naproxen; MITT Population; Test type: Superiority or Other; p = 0.0041, Regression, Cox; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.32 to 0.81]
Statistical Analysis 5: Comparison: Celecoxib vs Ibuprofen; MITT Population; Test type: Superiority or Other; p = 0.0003, Regression, Cox; Hazard Ratio (HR) = 0.43, 95% CI 2-sided [0.27 to 0.68]
Statistical Analysis 6: Comparison: Ibuprofen vs Naproxen; MITT Population; Test type: Superiority or Other; p = 0.4243, Regression, Cox; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.80 to 1.69]

4. Secondary Outcome: Change From Baseline in Patient's Assessment of Arthritis Pain (VAS)
Description: VAS question "How much pain do you have" was graded on a scale from 0 to 100 with 0 indicating "No pain" and 100 indicating "Worst possible pain".
Time Frame: ITT and MITT Population - Baseline to 42 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of participants
Arm/Group | Celecoxib | Ibuprofen | Naproxen
Number analyzed (Participants) | 8072 | 8040 | 7969
Number of participants
  Baseline (ITT) N= 8014, 8001, 7928 | 54.0 (23.53) | 54.1 (23.58) | 54.1 (24.04)
  Change-Baseline to Mon1 (ITT) N=7382, 7379, 7325 | -8.2 (24.69) | -9.0 (25.69) | -9.9 (25.53)
  Change-Baseline to Mon2 (ITT) N=7180, 7090, 7149 | -10.5 (26.39) | -10.6 (26.92) | -11.1 (26.83)
  Change-Baseline to Mon4 (ITT) N=6777, 6696, 6740 | -11.4 (27.70) | -11.7 (28.10) | -12.3 (27.80)
  Change-Baseline to Mon8 (ITT) N=6230, 6137, 6159 | -11.7 (28.92) | -12.1 (28.97) | -12.1 (28.83)
  Change-Baseline to Mon12 (ITT) N=5792, 5696, 5846 | -11.0 (29.15) | -11.6 (29.29) | -11.9 (29.30)
  Change-Baseline to Mon18 (ITT) N=5310, 5181. 5246 | -11.3 (29.11) | -11.3 (29.10) | -11.7 (29.33)
  Change-Baseline to Mon24 (ITT) N=4818, 4776, 4785 | -11.3 (29.44) | -11.5 (28.98) | -11.4 (29.27)
  Change-Baseline to Mon30 (ITT) N=4140, 4069, 4086 | -10.5 (29.81) | -11.2 (29.71) | -11.3 (29.71)
  Change-Baseline to Mon36 (ITT) N=3692, 3627, 3635 | -10.1 (29.61) | -10.7 (29.62) | -11.6 (29.80)
  Change-Baseline to Mon42 (ITT) N=3469, 3406, 3439 | -11.4 (29.78) | -11.1 (30.14) | -12.1 (30.27)
  Baseline (MITT) N=7974, 7954, 7894 | 54.0 (23.53) | 54.1 (23.58) | 54.1 (24.02)
  Change-Baseline to Mon1 MITT N=7372, 7367, 7321 | -8.2 (24.69) | -9.0 (25.67) | -9.9 (25.53)
  Change-Baseline to Mon2 MITT N=7170, 7078, 7142 | -10.5 (26.38) | -10.6 (26.92) | -11.1 (26.84)
  Change-Baseline to Mon4 MITT N=6772, 6686, 6732 | -11.4 (27.70) | -11.7 (28.10) | -12.3 (27.81)
  Change-Baseline to Mon8 MITT N=6224, 6128, 6155 | -11.7 (28.93) | -12.1 (28.97) | -12.1 (28.84)
  Change-Baseline to Mon12 MITT N=5787, 5689, 5844 | -11.0 (29.16) | -11.6 (29.30) | -11.9 (29.30)
  Change-Baseline to Mon18 MITT N=5305, 5175, 5242 | -11.3 (29.11) | -11.3 (29.12) | -11.7 (29.33)
  Change-Baseline to Mon24 MITT N=4815, 4769, 4782 | -11.4 (29.44) | -11.5 (29.00) | -11.3 (29.26)
  Change-Baseline to Mon30 MITT N=4139, 4067, 4085 | -10.5 (29.81) | -11.2 (29.71) | -11.3 (29.70)
  Change-Baseline to Mon36 MITT N=3691, 3623, 3635 | -10.2 (29.61) | -10.7 (29.62) | -11.6 (29.80)
  Change-Baseline to Mon42 MITT N=3468, 3404, 3438 | -11.4 (29.78) | -11.1 (30.14) | -12.1 (30.27)
Statistical Analysis 1: Comparison: Celecoxib vs Naproxen; Change from baseline to Month 1 (ITT); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 1.77, 95% CI 2-sided [1.01 to 2.53], Standard Error of Mean 0.39
Statistical Analysis 2: Comparison: Celecoxib vs Ibuprofen; Change from baseline to Month 1 (ITT); Test type: Superiority or Other; p = 0.0373, Mixed Models Analysis; Mean Difference (Final Values) = 0.81, 95% CI 2-sided [0.05 to 1.56], Standard Error of Mean 0.39
Statistical Analysis 3: Comparison: Ibuprofen vs Naproxen; Change from baseline to Month 1 (ITT); Test type: Superiority or Other; p = 0.0129, Mixed Models Analysis; Mean Difference (Final Values) = 0.96, 95% CI 2-sided [0.20 to 1.72], Standard Error of Mean 0.39
Statistical Analysis 4: Comparison: Celecoxib vs Naproxen; Change from baseline to Month 2 (ITT); Test type: Superiority or Other; p = 0.1830, Mixed Models Analysis; Mean Difference (Final Values) = 0.52, 95% CI 2-sided [-0.25 to 1.29], Standard Error of Mean 0.39
Statistical Analysis 5: Comparison: Celecoxib vs Ibuprofen; Change from baseline to Month 2 (ITT); Test type: Superiority or Other; p = 0.7777, Mixed Models Analysis; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.88 to 0.66], Standard Error of Mean 0.39
Statistical Analysis 6: Comparison: Ibuprofen vs Naproxen; Change from baseline to Month 2 (ITT); Test type: Superiority or Other; p = 0.1072, Mixed Models Analysis; Mean Difference (Final Values) = 0.63, 95% CI 2-sided [-0.14 to 1.40], Standard Error of Mean 0.39
Statistical Analysis 7: Comparison: Celecoxib vs Naproxen; Change from baseline to Month 4 (ITT); Test type: Superiority or Other; p = 0.8237, Mixed Models Analysis; Mean Difference (Final Values) = 0.67, 95% CI 2-sided [-0.12 to 1.46], Standard Error of Mean 0.40
Statistical Analysis 8: Comparison: Celecoxib vs Ibuprofen; Change from baseline to Month 4 (ITT); Test type: Superiority or Other; p = 0.8237, Mixed Models Analysis; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.88 to 0.70], Standard Error of Mean 0.40
Statistical Analysis 9: Comparison: Ibuprofen vs Naproxen; Change from baseline to Month 4 (ITT); Test type: Superiority or Other; p = 0.0587, Mixed Models Analysis; Mean Difference (Final Values) = 0.76, 95% CI 2-sided [-0.03 to 1.55], Standard Error of Mean 0.40
Statistical Analysis 10: Comparison: Celecoxib vs Naproxen; Change from baseline to Month 8 (ITT); Test type: Superiority or Other; p = 0.3129, Mixed Models Analysis; Mean Difference (Final Values) = 0.42, 95% CI 2-sided [-0.39 to 1.23], Standard Error of Mean 0.41
Statistical Analysis 11: Comparison: Celecoxib vs Ibuprofen; Change from baseline to Month 8 (ITT); Test type: Superiority or Other; p = 0.6526, Mixed Models Analysis; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-0.63 to 1.00], Standard Error of Mean 0.41
Statistical Analysis 12: Comparison: Ibuprofen vs Naproxen; Change from baseline to Month 8 (ITT); Test type: Superiority or Other; p = 0.5774, Mixed Models Analysis; Mean Difference (Final Values) = 0.23, 95% CI 2-sided [-0.58 to 1.05], Standard Error of Mean 0.42
Statistical Analysis 13: Comparison: Celecoxib vs Naproxen; Change from baseline to Month 12 (ITT); Test type: Superiority or Other; p = 0.0632, Mixed Models Analysis; Mean Difference (Final Values) = 0.79, 95% CI 2-sided [-0.04 to 1.62], Standard Error of Mean 0.42
Statistical Analysis 14: Comparison: Celecoxib vs Ibuprofen; Change from baseline to Month 12 (ITT); Test type: Superiority or Other; p = 0.4540, Mixed Models Analysis; Mean Difference (Final Values) = 0.32, 95% CI 2-sided [-0.52 to 1.15], Standard Error of Mean 0.43
Statistical Analysis 15: Comparison: Ibuprofen vs Naproxen; Change from baseline to Month 12 (ITT); Test type: Superiority or Other; p = 0.2705, Mixed Models Analysis; Mean Difference (Final Values) = 0.47, 95% CI 2-sided [-0.37 to 1.30], Standard Error of Mean 0.43
Statistical Analysis 16: Comparison: Celecoxib vs Naproxen; Change from baseline to Month 18 (ITT); Test type: Superiority or Other; p = 0.5225, Mixed Models Analysis; Mean Difference (Final Values) = 0.28, 95% CI 2-sided [-0.58 to 1.14], Standard Error of Mean 0.44
Statistical Analysis 17: Comparison: Celecoxib vs Ibuprofen; Change from baseline to Month 18 (ITT); Test type: Superiority or Other; p = 0.5996, Mixed Models Analysis; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-1.10 to 0.63], Standard Error of Mean 0.44
Statistical Analysis 18: Comparison: Ibuprofen vs Naproxen; Change from baseline to Month 18 (ITT); Test type: Superiority or Other; p = 0.2461, Mixed Models Analysis; Mean Difference (Final Values) = 0.51, 95% CI 2-sided [-0.35 to 1.38], Standard Error of Mean 0.44
Statistical Analysis 19: Comparison: Celecoxib vs Naproxen; Change from baseline to Month 24 (ITT); Test type: Superiority or Other; p = 0.8127, Mixed Models Analysis; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.79 to 1.00], Standard Error of Mean 0.46
Statistical Analysis 20: Comparison: Celecoxib vs Ibuprofen; Change from baseline to Month 24 (ITT); Test type: Superiority or Other; p = 0.9641, Mixed Models Analysis; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.92 to 0.87], Standard Error of Mean 0.46
Statistical Analysis 21: Comparison: Ibuprofen vs Naproxen; Change from baseline to Month 24 (ITT); Test type: Superiority or Other; p = 0.7784, Mixed Models Analysis; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-0.77 to 1.03], Standard Error of Mean 0.46
Statistical Analysis 22: Comparison: Celecoxib vs Naproxen; Change from baseline to Month 30 (ITT); Test type: Superiority or Other; p = 0.2105, Mixed Models Analysis; Mean Difference (Final Values) = 0.61, 95% CI 2-sided [-0.34 to 1.56], Standard Error of Mean 0.49
Statistical Analysis 23: Comparison: Celecoxib vs Ibuprofen; Change from baseline to Month 30 (ITT); Test type: Superiority or Other; p = 0.2909, Mixed Models Analysis; Mean Difference (Final Values) = 0.51, 95% CI 2-sided [-0.44 to 1.46], Standard Error of Mean 0.49
Statistical Analysis 24: Comparison: Ibuprofen vs Naproxen; Change from baseline to Month 30 (ITT); Test type: Superiority or Other; p = 0.8459, Mixed Models Analysis; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-0.86 to 1.05], Standard Error of Mean 0.49
Statistical Analysis 25: Comparison: Celecoxib vs Naproxen; Change from baseline to Month 36 (ITT); Test type: Superiority or Other; p = 0.1116, Mixed Models Analysis; Mean Difference (Final Values) = 0.81, 95% CI 2-sided [-0.19 to 1.80], Standard Error of Mean 0.51
Statistical Analysis 26: Comparison: Celecoxib vs Ibuprofen; Change from baseline to Month 36 (ITT); Test type: Superiority or Other; p = 0.9751, Mixed Models Analysis; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.98 to 1.01], Standard Error of Mean 0.51
Statistical Analysis 27: Comparison: Ibuprofen vs Naproxen; Change from baseline to Month 36 (ITT); Test type: Superiority or Other; p = 0.1202, Mixed Models Analysis; Mean Difference (Final Values) = 0.79, 95% CI 2-sided [-0.21 to 1.79], Standard Error of Mean 0.51
Statistical Analysis 28: Comparison: Celecoxib vs Naproxen; Change from baseline to Month 42 (ITT); Test type: Superiority or Other; p = 0.3767, Mixed Models Analysis; Mean Difference (Final Values) = 0.46, 95% CI 2-sided [-0.56 to 1.48], Standard Error of Mean 0.52
Statistical Analysis 29: Comparison: Celecoxib vs Ibuprofen; Change from baseline to Month 42 (ITT); Test type: Superiority or Other; p = 0.1123, Mixed Models Analysis; Mean Difference (Final Values) = -0.83, 95% CI 2-sided [-1.85 to 0.19], Standard Error of Mean 0.52
Statistical Analysis 30: Comparison: Ibuprofen vs Naproxen; Change from baseline to Month 42 (ITT); Test type: Superiority or Other; p = 0.0137, Mixed Models Analysis; Mean Difference (Final Values) = 1.29, 95% CI 2-sided [0.26 to 2.31], Standard Error of Mean 0.52
Statistical Analysis 31: Comparison: Celecoxib vs Naproxen; Change from Baseline to Month 1 (MITT); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 1.77, 95% CI 2-sided [1.07 to 2.47], Standard Error of Mean 0.36
Statistical Analysis 32: Comparison: Celecoxib vs Ibuprofen; Change from Baseline to Month 1 (MITT); Test type: Superiority or Other; p = 0.0197, Mixed Models Analysis; Mean Difference (Final Values) = 0.84, 95% CI 2-sided [0.13 to 1.54], Standard Error of Mean 0.36
Statistical Analysis 33: Comparison: Ibuprofen vs Naproxen; Change from Baseline to Month 1 (MITT); Test type: Superiority or Other; p = 0.0094, Mixed Models Analysis; Mean Difference (Final Values) = 0.93, 95% CI 2-sided [0.23 to 1.64], Standard Error of Mean 0.36
Statistical Analysis 34: Comparison: Celecoxib vs Naproxen; Change from baseline to Month 2 (MITT); Test type: Superiority or Other; p = 0.1247, Mixed Models Analysis; Mean Difference (Final Values) = 0.57, 95% CI 2-sided [-0.16 to 1.31], Standard Error of Mean 0.37
Statistical Analysis 35: Comparison: Celecoxib vs Ibuprofen; Change from baseline to Month 2 (MITT); Test type: Superiority or Other; p = 0.8278, Mixed Models Analysis; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.81 to 0.65], Standard Error of Mean 0.37
Statistical Analysis 36: Comparison: Ibuprofen vs Naproxen; Change from baseline to Month 2 (MITT); Test type: Superiority or Other; p = 0.0802, Mixed Models Analysis; Mean Difference (Final Values) = 0.65, 95% CI 2-sided [-0.08 to 1.39], Standard Error of Mean 0.37
Statistical Analysis 37: Comparison: Celecoxib vs Naproxen; Change from baseline to Month 4 (MITT); Test type: Superiority or Other; p = 0.0822, Mixed Models Analysis; Mean Difference (Final Values) = 0.68, 95% CI 2-sided [-0.09 to 1.46], Standard Error of Mean 0.39
Statistical Analysis 38: Comparison: Celecoxib vs Ibuprofen; Change from baseline to Month 4 (MITT); Test type: Superiority or Other; p = 0.8314, Mixed Models Analysis; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.86 to 0.69], Standard Error of Mean 0.39
Statistical Analysis 39: Comparison: Ibuprofen vs Naproxen; Change from baseline to Month 4 (MITT); Test type: Superiority or Other; p = 0.0516, Mixed Models Analysis; Mean Difference (Final Values) = 0.77, 95% CI 2-sided [-0.01 to 1.54], Standard Error of Mean 0.39
Statistical Analysis 40: Comparison: Celecoxib vs Naproxen; Change from baseline to Month 8 (MITT); Test type: Superiority or Other; p = 0.3202, Mixed Models Analysis; Mean Difference (Final Values) = 0.42, 95% CI 2-sided [-0.40 to 1.24], Standard Error of Mean 0.42
Statistical Analysis 41: Comparison: Celecoxib vs Ibuprofen; Change from baseline to Month 8 (MITT); Test type: Superiority or Other; p = 0.5893, Mixed Models Analysis; Mean Difference (Final Values) = 0.23, 95% CI 2-sided [-0.60 to 1.05], Standard Error of Mean 0.42
Statistical Analysis 42: Comparison: Ibuprofen vs Naproxen; Change from baseline to Month 8 (MITT); Test type: Superiority or Other; p = 0.6510, Mixed Models Analysis; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-0.63 to 1.01], Standard Error of Mean 0.42
Statistical Analysis 43: Comparison: Celecoxib vs Naproxen; Change from baseline to Month 12 (MITT); Test type: Superiority or Other; p = 0.0796, Mixed Models Analysis; Mean Difference (Final Values) = 0.76, 95% CI 2-sided [-0.09 to 1.62], Standard Error of Mean 0.44
Statistical Analysis 44: Comparison: Celecoxib vs Ibuprofen; Change from baseline to Month 12 (MITT); Test type: Superiority or Other; p = 0.5061, Mixed Models Analysis; Mean Difference (Final Values) = 0.29, 95% CI 2-sided [-0.57 to 1.15], Standard Error of Mean 0.44
Statistical Analysis 45: Comparison: Ibuprofen vs Naproxen; Change from baseline to Month 12 (MITT); Test type: Superiority or Other; p = 0.2796, Mixed Models Analysis; Mean Difference (Final Values) = 0.47, 95% CI 2-sided [-0.38 to 1.33], Standard Error of Mean 0.44
Statistical Analysis 46: Comparison: Celecoxib vs Naproxen; Change from baseline to Month 18 (MITT); Test type: Superiority or Other; p = 0.6725, Mixed Models Analysis; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-0.69 to 1.08], Standard Error of Mean 0.45
Statistical Analysis 47: Comparison: Celecoxib vs Ibuprofen; Change from baseline to Month 18 (MITT); Test type: Superiority or Other; p = 0.6381, Mixed Models Analysis; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-1.10 to 0.67], Standard Error of Mean 0.45
Statistical Analysis 48: Comparison: Ibuprofen vs Naproxen; Change from baseline to Month 18 (MITT); Test type: Superiority or Other; p = 0.3737, Mixed Models Analysis; Mean Difference (Final Values) = 0.40, 95% CI 2-sided [-0.49 to 1.29], Standard Error of Mean 0.45
Statistical Analysis 49: Comparison: Celecoxib vs Naproxen; Change from baseline to Month 24 (MITT); Test type: Superiority or Other; p = 0.9139, Mixed Models Analysis; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.87 to 0.97], Standard Error of Mean 0.47
Statistical Analysis 50: Comparison: Celecoxib vs Ibuprofen; Change from baseline to Month 24 (MITT); Test type: Superiority or Other; p = 0.9998, Mixed Models Analysis; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.92 to 0.92], Standard Error of Mean 0.47
Statistical Analysis 51: Comparison: Ibuprofen vs Naproxen; Change from baseline to Month 24 (MITT); Test type: Superiority or Other; p = 0.9144, Mixed Models Analysis; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.88 to 0.98], Standard Error of Mean 0.47
Statistical Analysis 52: Comparison: Celecoxib vs Naproxen; Change from baseline to Month 30 (MITT); Test type: Superiority or Other; p = 0.2250, Mixed Models Analysis; Mean Difference (Final Values) = 0.62, 95% CI 2-sided [-0.38 to 1.61], Standard Error of Mean 0.51
Statistical Analysis 53: Comparison: Celecoxib vs Ibuprofen; Change from baseline to Month 30 (MITT); Test type: Superiority or Other; p = 0.2758, Mixed Models Analysis; Mean Difference (Final Values) = 0.55, 95% CI 2-sided [-0.44 to 1.55], Standard Error of Mean 0.51
Statistical Analysis 54: Comparison: Ibuprofen vs Naproxen; Change from baseline to Month 30 (MITT); Test type: Superiority or Other; p = 0.9030, Mixed Models Analysis; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.94 to 1.06], Standard Error of Mean 0.51
Statistical Analysis 55: Comparison: Celecoxib vs Naproxen; Change from baseline to Month 36 (MITT); Test type: Superiority or Other; p = 0.0910, Mixed Models Analysis; Mean Difference (Final Values) = 0.90, 95% CI 2-sided [-0.14 to 1.94], Standard Error of Mean 0.53
Statistical Analysis 56: Comparison: Celecoxib vs Ibuprofen; Change from baseline to Month 36 (MITT); Test type: Superiority or Other; p = 0.7668, Mixed Models Analysis; Mean Difference (Final Values) = 0.16, 95% CI 2-sided [-0.88 to 1.20], Standard Error of Mean 0.53
Statistical Analysis 57: Comparison: Ibuprofen vs Naproxen; Change from baseline to Month 36 (MITT); Test type: Superiority or Other; p = 0.1653, Mixed Models Analysis; Mean Difference (Final Values) = 0.74, 95% CI 2-sided [-0.31 to 1.78], Standard Error of Mean 0.53
Statistical Analysis 58: Comparison: Celecoxib vs Naproxen; Change from baseline to Month 42 (MITT); Test type: Superiority or Other; p = 0.4323, Mixed Models Analysis; Mean Difference (Final Values) = 0.43, 95% CI 2-sided [-0.65 to 1.52], Standard Error of Mean 0.55
Statistical Analysis 59: Comparison: Celecoxib vs Ibuprofen; Change from baseline to Month 42 (MITT); Test type: Superiority or Other; p = 0.1439, Mixed Models Analysis; Mean Difference (Final Values) = -0.81, 95% CI 2-sided [-1.89 to 0.28], Standard Error of Mean 0.55
Statistical Analysis 60: Comparison: Ibuprofen vs Naproxen; Change from baseline to Month 42 (MITT); Test type: Superiority or Other; p = 0.0251, Mixed Models Analysis; Mean Difference (Final Values) = 1.24, 95% CI 2-sided [0.16 to 2.33], Standard Error of Mean 0.55

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the signing of the informed consent throughout the entire study period (42 months) and including 30 calendar days after the last administration of the investigational product.
Arm/Group | Celecoxib | Ibuprofen | Naproxen
Serious Adverse Events (participants affected / at risk) | 1473/8030 | 1624/7992 | 1611/7933
Other Adverse Events (participants affected / at risk) | 4268/8030 | 4363/7992 | 4337/7933
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Celecoxib (N=8030) | Ibuprofen (N=7992) | Naproxen (N=7933)
Anaemia (Blood and lymphatic system disorders) | 15 | 34 | 24
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 0 | 1 | 0
Aplastic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Coagulopathy (Blood and lymphatic system disorders) | 1 | 1 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 2 | 1 | 2
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 10 | 11
Leukocytosis (Blood and lymphatic system disorders) | 1 | 2 | 5
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 | 1 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 3
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 7 | 7 | 3
Acute left ventricular failure (Cardiac disorders) | 1 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 22 | 20 | 18
Angina pectoris (Cardiac disorders) | 13 | 11 | 13
Angina unstable (Cardiac disorders) | 45 | 41 | 60
Aortic valve disease (Cardiac disorders) | 0 | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 0 | 2 | 3
Aortic valve stenosis (Cardiac disorders) | 3 | 1 | 2
Arrhythmia (Cardiac disorders) | 1 | 7 | 3
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 5 | 5 | 7
Arteriospasm coronary (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 35 | 39 | 36
Atrial flutter (Cardiac disorders) | 6 | 4 | 4
Atrioventricular block (Cardiac disorders) | 1 | 3 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 7 | 2
Atrioventricular block second degree (Cardiac disorders) | 2 | 2 | 3
Atrioventricular dissociation (Cardiac disorders) | 0 | 1 | 0
Bradyarrhythmia (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 10 | 11 | 6
Bundle branch block left (Cardiac disorders) | 0 | 1 | 1
Bundle branch block right (Cardiac disorders) | 0 | 0 | 1
Cardiac aneurysm (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 6 | 9 | 6
Cardiac disorder (Cardiac disorders) | 1 | 2 | 0
Cardiac failure (Cardiac disorders) | 2 | 8 | 4
Cardiac failure chronic (Cardiac disorders) | 1 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 31 | 41 | 41
Cardiac tamponade (Cardiac disorders) | 0 | 1 | 0
Cardiac valve disease (Cardiac disorders) | 1 | 0 | 1
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 6 | 5 | 4
Cardiogenic shock (Cardiac disorders) | 0 | 3 | 2
Cardiomyopathy (Cardiac disorders) | 3 | 4 | 2
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 | 0
Cardiovascular disorder (Cardiac disorders) | 0 | 1 | 2
Congestive cardiomyopathy (Cardiac disorders) | 1 | 1 | 1
Cor pulmonale chronic (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 42 | 40 | 44
Coronary artery insufficiency (Cardiac disorders) | 1 | 2 | 1
Coronary artery occlusion (Cardiac disorders) | 9 | 8 | 8
Coronary artery stenosis (Cardiac disorders) | 4 | 9 | 6
Coronary artery thrombosis (Cardiac disorders) | 0 | 1 | 0
Extrasystoles (Cardiac disorders) | 2 | 0 | 0
Heart valve incompetence (Cardiac disorders) | 1 | 0 | 0
Hypertensive cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Hypertensive heart disease (Cardiac disorders) | 0 | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 3 | 0 | 3
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 1
Left ventricular failure (Cardiac disorders) | 2 | 0 | 0
Mitral valve disease (Cardiac disorders) | 1 | 1 | 1
Mitral valve incompetence (Cardiac disorders) | 2 | 2 | 0
Myocardial infarction (Cardiac disorders) | 45 | 70 | 48
Myocardial ischaemia (Cardiac disorders) | 2 | 7 | 3
Nodal arrhythmia (Cardiac disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 2 | 3 | 4
Pericardial effusion (Cardiac disorders) | 1 | 2 | 1
Pericarditis (Cardiac disorders) | 0 | 1 | 4
Pleuropericarditis (Cardiac disorders) | 0 | 1 | 0
Postinfarction angina (Cardiac disorders) | 1 | 0 | 0
Prinzmetal angina (Cardiac disorders) | 2 | 0 | 0
Silent myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 3 | 3
Sinus node dysfunction (Cardiac disorders) | 2 | 3 | 4
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 8 | 4
Tachyarrhythmia (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 2 | 2 | 5
Tricuspid valve incompetence (Cardiac disorders) | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 3 | 3
Ventricular fibrillation (Cardiac disorders) | 0 | 2 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 2
Arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 0 | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 2
Cardiac septal defect (Congenital, familial and genetic disorders) | 1 | 0 | 0
Cerebrovascular arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 0 | 1
Choledochal cyst (Congenital, familial and genetic disorders) | 0 | 1 | 0
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 0 | 1 | 0
Diverticulitis Meckel's (Congenital, familial and genetic disorders) | 0 | 1 | 0
Haemorrhagic arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 1 | 1
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 | 3 | 0
Renal hypoplasia (Congenital, familial and genetic disorders) | 0 | 0 | 1
Deafness (Ear and labyrinth disorders) | 1 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 5 | 2 | 8
Vertigo positional (Ear and labyrinth disorders) | 0 | 3 | 3
Adrenal haemorrhage (Endocrine disorders) | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 2 | 0 | 0
Autoimmune thyroiditis (Endocrine disorders) | 1 | 0 | 0
Goitre (Endocrine disorders) | 2 | 4 | 0
Hyperparathyroidism (Endocrine disorders) | 3 | 4 | 0
Hyperparathyroidism primary (Endocrine disorders) | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0
Hypogonadism (Endocrine disorders) | 1 | 0 | 0
Hypoparathyroidism (Endocrine disorders) | 0 | 0 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 1
Myxoedema (Endocrine disorders) | 0 | 0 | 1
Parathyroid disorder (Endocrine disorders) | 0 | 1 | 0
Thyroid mass (Endocrine disorders) | 2 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 1 | 1
Eye haemorrhage (Eye disorders) | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 2 | 0
Optic neuropathy (Eye disorders) | 0 | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0 | 0
Retinal haemorrhage (Eye disorders) | 1 | 1 | 0
Retinal vein occlusion (Eye disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 2
Visual impairment (Eye disorders) | 0 | 0 | 1
Vitreous detachment (Eye disorders) | 1 | 0 | 0
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal hernia (Gastrointestinal disorders) | 5 | 4 | 7
Abdominal incarcerated hernia (Gastrointestinal disorders) | 3 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 14 | 7 | 13
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 3 | 2
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 2 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
Autoimmune pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Chronic gastritis (Gastrointestinal disorders) | 0 | 2 | 0
Colitis (Gastrointestinal disorders) | 6 | 3 | 3
Colitis ischaemic (Gastrointestinal disorders) | 1 | 4 | 4
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 1
Colonic fistula (Gastrointestinal disorders) | 1 | 0 | 0
Colonic pseudo-obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 3 | 1
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 8 | 5
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 0 | 3 | 1
Diverticulum (Gastrointestinal disorders) | 6 | 0 | 2
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 2 | 2
Duodenal ulcer (Gastrointestinal disorders) | 2 | 2 | 3
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 2
Duodenitis (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 1
Enteritis (Gastrointestinal disorders) | 1 | 1 | 0
Enterocele (Gastrointestinal disorders) | 0 | 0 | 2
Enterovesical fistula (Gastrointestinal disorders) | 0 | 0 | 1
Erosive duodenitis (Gastrointestinal disorders) | 0 | 0 | 2
Erosive oesophagitis (Gastrointestinal disorders) | 1 | 2 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1 | 2
Femoral hernia (Gastrointestinal disorders) | 0 | 1 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 12 | 5
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0
Gastric varices (Gastrointestinal disorders) | 0 | 1 | 0
Gastric varices haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Gastric volvulus (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 3 | 6 | 5
Gastritis erosive (Gastrointestinal disorders) | 1 | 6 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 2
Gastroduodenal haemorrhage (Gastrointestinal disorders) | 0 | 3 | 2
Gastroduodenitis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 7 | 8 | 8
Gastrointestinal hypomotility (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal stenosis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal ulcer (Gastrointestinal disorders) | 1 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 3 | 4
Haematochezia (Gastrointestinal disorders) | 0 | 2 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1
Hernial eventration (Gastrointestinal disorders) | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 2 | 2 | 2
Ileal ulcer (Gastrointestinal disorders) | 2 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 3 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 0 | 1
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1
Inflammatory bowel disease (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 5 | 2 | 0
Intestinal dilatation (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 2
Intestinal obstruction (Gastrointestinal disorders) | 2 | 2 | 5
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 3
Intestinal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0 | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 4 | 3 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Large intestinal ulcer (Gastrointestinal disorders) | 1 | 2 | 2
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 2
Large intestine polyp (Gastrointestinal disorders) | 1 | 2 | 0
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 0 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 3 | 3
Megacolon (Gastrointestinal disorders) | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 1
Mesenteric artery stenosis (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 3 | 6
Necrotising colitis (Gastrointestinal disorders) | 1 | 0 | 0
Neutropenic colitis (Gastrointestinal disorders) | 0 | 1 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 1 | 1
Oedematous pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Oesophageal spasm (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 2 | 2
Oesophagitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatic cyst (Gastrointestinal disorders) | 1 | 0 | 1
Pancreatic necrosis (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 8 | 12 | 12
Pancreatitis acute (Gastrointestinal disorders) | 3 | 4 | 6
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1 | 1
Pancreatitis necrotising (Gastrointestinal disorders) | 0 | 1 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 4 | 4 | 2
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 0 | 1
Retroperitoneal mass (Gastrointestinal disorders) | 0 | 1 | 0
Salivary gland calculus (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 7 | 9 | 8
Umbilical hernia (Gastrointestinal disorders) | 4 | 0 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2 | 1
Volvulus (Gastrointestinal disorders) | 0 | 3 | 0
Vomiting (Gastrointestinal disorders) | 5 | 7 | 7
Adverse drug reaction (General disorders) | 0 | 0 | 1
Asthenia (General disorders) | 4 | 5 | 4
Cardiac death (General disorders) | 0 | 1 | 0
Chest discomfort (General disorders) | 2 | 5 | 4
Chest pain (General disorders) | 52 | 84 | 73
Complication associated with device (General disorders) | 1 | 0 | 2
Cyst rupture (General disorders) | 0 | 0 | 1
Death (General disorders) | 4 | 3 | 7
Device related thrombosis (General disorders) | 0 | 0 | 1
Drowning (General disorders) | 0 | 0 | 1
Drug interaction (General disorders) | 0 | 0 | 1
Electrocution (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 2 | 2 | 2
Feeling hot (General disorders) | 0 | 1 | 0
General physical health deterioration (General disorders) | 1 | 1 | 0
Generalised oedema (General disorders) | 0 | 1 | 1
Granuloma (General disorders) | 0 | 0 | 1
Hernia (General disorders) | 0 | 3 | 1
Ill-defined disorder (General disorders) | 0 | 0 | 1
Impaired healing (General disorders) | 1 | 1 | 2
Incarcerated hernia (General disorders) | 1 | 1 | 0
Influenza like illness (General disorders) | 0 | 1 | 0
Local swelling (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 0 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 1
Necrosis (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 23 | 19 | 23
Oedema peripheral (General disorders) | 4 | 1 | 1
Organ failure (General disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 1
Pelvic mass (General disorders) | 0 | 1 | 1
Peripheral swelling (General disorders) | 1 | 0 | 2
Polyp (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 4 | 3
Sudden cardiac death (General disorders) | 0 | 0 | 1
Sudden death (General disorders) | 0 | 1 | 0
Surgical failure (General disorders) | 0 | 1 | 2
Systemic inflammatory response syndrome (General disorders) | 0 | 1 | 0
Vascular stent stenosis (General disorders) | 0 | 1 | 0
Vascular stent thrombosis (General disorders) | 1 | 0 | 0
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 2 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 5
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 1
Biliary dyskinesia (Hepatobiliary disorders) | 1 | 1 | 1
Biliary tract disorder (Hepatobiliary disorders) | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 8 | 10 | 11
Cholecystitis acute (Hepatobiliary disorders) | 9 | 11 | 5
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 3
Cholelithiasis (Hepatobiliary disorders) | 24 | 23 | 12
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 1 | 0
Gallbladder disorder (Hepatobiliary disorders) | 0 | 1 | 1
Hepatic cyst (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic lesion (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic vein thrombosis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatitis alcoholic (Hepatobiliary disorders) | 1 | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1 | 0
Jaundice hepatocellular (Hepatobiliary disorders) | 0 | 0 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 1
Allergy to arthropod bite (Immune system disorders) | 0 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 2
Anaphylactic shock (Immune system disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 3
Hypersensitivity (Immune system disorders) | 1 | 2 | 1
Sarcoidosis (Immune system disorders) | 1 | 0 | 0
Abdominal abscess (Infections and infestations) | 1 | 1 | 1
Abdominal infection (Infections and infestations) | 1 | 0 | 0
Abdominal wall abscess (Infections and infestations) | 1 | 1 | 0
Abscess intestinal (Infections and infestations) | 0 | 0 | 1
Abscess limb (Infections and infestations) | 2 | 3 | 2
Abscess neck (Infections and infestations) | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 1 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 0
Appendiceal abscess (Infections and infestations) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 7 | 7 | 7
Appendicitis perforated (Infections and infestations) | 2 | 3 | 2
Arthritis bacterial (Infections and infestations) | 5 | 2 | 2
Arthritis infective (Infections and infestations) | 0 | 2 | 3
Atypical pneumonia (Infections and infestations) | 0 | 0 | 2
Bacteraemia (Infections and infestations) | 1 | 1 | 0
Bacterial diarrhoea (Infections and infestations) | 1 | 0 | 1
Bacterial disease carrier (Infections and infestations) | 0 | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 2 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 1
Beta haemolytic streptococcal infection (Infections and infestations) | 0 | 1 | 0
Bone tuberculosis (Infections and infestations) | 0 | 0 | 1
Breast abscess (Infections and infestations) | 0 | 1 | 1
Bronchitis (Infections and infestations) | 10 | 16 | 17
Bronchitis bacterial (Infections and infestations) | 1 | 1 | 0
Bursitis infective (Infections and infestations) | 2 | 0 | 1
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 29 | 32 | 32
Cellulitis of male external genital organ (Infections and infestations) | 0 | 0 | 1
Cellulitis staphylococcal (Infections and infestations) | 1 | 1 | 2
Cholecystitis infective (Infections and infestations) | 0 | 2 | 1
Chronic pulmonary histoplasmosis (Infections and infestations) | 1 | 0 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 2 | 4 | 4
Clostridium difficile infection (Infections and infestations) | 1 | 2 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 1 | 0
Dengue fever (Infections and infestations) | 0 | 1 | 1
Device related infection (Infections and infestations) | 1 | 4 | 3
Diabetic foot infection (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 12 | 13 | 17
Embolic pneumonia (Infections and infestations) | 0 | 0 | 1
Empyema (Infections and infestations) | 1 | 1 | 1
Encephalitis (Infections and infestations) | 0 | 1 | 0
Endocarditis (Infections and infestations) | 0 | 1 | 0
Epididymitis (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 1 | 2 | 2
Escherichia bacteraemia (Infections and infestations) | 1 | 0 | 1
Escherichia infection (Infections and infestations) | 1 | 0 | 0
Escherichia sepsis (Infections and infestations) | 1 | 1 | 2
Escherichia urinary tract infection (Infections and infestations) | 2 | 1 | 0
Extradural abscess (Infections and infestations) | 2 | 2 | 0
Gangrene (Infections and infestations) | 1 | 1 | 1
Gastroenteritis (Infections and infestations) | 12 | 21 | 7
Gastroenteritis bacterial (Infections and infestations) | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 4 | 4 | 3
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0
Gastrointestinal viral infection (Infections and infestations) | 1 | 0 | 0
Genitourinary tract infection (Infections and infestations) | 0 | 0 | 1
Groin abscess (Infections and infestations) | 1 | 0 | 1
H1N1 influenza (Infections and infestations) | 1 | 0 | 0
HIV infection (Infections and infestations) | 0 | 0 | 1
Haemophilus infection (Infections and infestations) | 1 | 0 | 0
Helicobacter gastritis (Infections and infestations) | 0 | 1 | 0
Hepatic infection (Infections and infestations) | 1 | 0 | 0
Herpes oesophagitis (Infections and infestations) | 1 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 1 | 0
Incision site infection (Infections and infestations) | 0 | 0 | 1
Infected skin ulcer (Infections and infestations) | 1 | 0 | 2
Infection (Infections and infestations) | 1 | 1 | 1
Infectious colitis (Infections and infestations) | 0 | 1 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 0 | 2
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 0 | 1
Infective tenosynovitis (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 2 | 4 | 1
Intervertebral discitis (Infections and infestations) | 1 | 1 | 2
Joint abscess (Infections and infestations) | 0 | 0 | 1
Kidney infection (Infections and infestations) | 1 | 1 | 1
Klebsiella bacteraemia (Infections and infestations) | 1 | 0 | 1
Klebsiella infection (Infections and infestations) | 1 | 0 | 0
Liver abscess (Infections and infestations) | 2 | 1 | 0
Localised infection (Infections and infestations) | 4 | 2 | 5
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 2
Lung infection (Infections and infestations) | 1 | 2 | 0
Lymphangitis (Infections and infestations) | 0 | 1 | 1
Meningitis bacterial (Infections and infestations) | 1 | 0 | 0
Meningitis pneumococcal (Infections and infestations) | 0 | 0 | 1
Necrotising fasciitis (Infections and infestations) | 0 | 2 | 1
Nosocomial infection (Infections and infestations) | 0 | 0 | 2
Ophthalmic herpes zoster (Infections and infestations) | 0 | 1 | 1
Oral candidiasis (Infections and infestations) | 1 | 0 | 0
Orchitis (Infections and infestations) | 0 | 1 | 1
Osteomyelitis (Infections and infestations) | 9 | 6 | 8
Osteomyelitis acute (Infections and infestations) | 1 | 0 | 3
Osteomyelitis chronic (Infections and infestations) | 1 | 0 | 0
Otitis media (Infections and infestations) | 0 | 1 | 0
Pancreatic abscess (Infections and infestations) | 1 | 0 | 0
Pancreatitis bacterial (Infections and infestations) | 1 | 0 | 0
Pancreatitis viral (Infections and infestations) | 0 | 1 | 0
Parametritis (Infections and infestations) | 0 | 1 | 0
Paraspinal abscess (Infections and infestations) | 1 | 0 | 0
Parotitis (Infections and infestations) | 0 | 1 | 0
Periodontitis (Infections and infestations) | 1 | 0 | 0
Perirectal abscess (Infections and infestations) | 0 | 1 | 0
Peritonitis (Infections and infestations) | 1 | 3 | 1
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 1
Peritonsillar abscess (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 1
Pleurisy viral (Infections and infestations) | 0 | 1 | 0
Pneumococcal sepsis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 64 | 79 | 69
Pneumonia bacterial (Infections and infestations) | 3 | 1 | 1
Pneumonia fungal (Infections and infestations) | 0 | 0 | 1
Pneumonia haemophilus (Infections and infestations) | 0 | 0 | 1
Pneumonia klebsiella (Infections and infestations) | 0 | 0 | 1
Pneumonia pseudomonal (Infections and infestations) | 0 | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 2 | 1 | 1
Pneumonia streptococcal (Infections and infestations) | 0 | 0 | 1
Post procedural infection (Infections and infestations) | 2 | 0 | 2
Postoperative abscess (Infections and infestations) | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 3 | 2 | 2
Prostate infection (Infections and infestations) | 1 | 0 | 0
Proteus infection (Infections and infestations) | 0 | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 1 | 0 | 1
Pyelonephritis (Infections and infestations) | 5 | 9 | 8
Pyelonephritis acute (Infections and infestations) | 5 | 3 | 3
Pyelonephritis chronic (Infections and infestations) | 0 | 1 | 0
Pyometra (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 3
Sepsis (Infections and infestations) | 19 | 20 | 12
Septic arthritis staphylococcal (Infections and infestations) | 1 | 0 | 3
Septic shock (Infections and infestations) | 2 | 5 | 4
Sinusitis (Infections and infestations) | 0 | 5 | 0
Skin infection (Infections and infestations) | 1 | 0 | 1
Spinal cord abscess (Infections and infestations) | 1 | 0 | 0
Staphylococcal abscess (Infections and infestations) | 1 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 2 | 1 | 0
Staphylococcal infection (Infections and infestations) | 4 | 2 | 4
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 2
Staphylococcal skin infection (Infections and infestations) | 0 | 0 | 1
Stenotrophomonas infection (Infections and infestations) | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 4 | 2 | 1
Tinea pedis (Infections and infestations) | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 2
Tooth abscess (Infections and infestations) | 0 | 2 | 2
Tooth infection (Infections and infestations) | 0 | 0 | 1
Tuberculosis (Infections and infestations) | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 1 | 1
Urinary tract infection (Infections and infestations) | 16 | 22 | 20
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 1
Urosepsis (Infections and infestations) | 9 | 8 | 6
Viral diarrhoea (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 1 | 2 | 3
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Vulval abscess (Infections and infestations) | 0 | 1 | 1
Wound infection (Infections and infestations) | 1 | 0 | 2
Wound infection staphylococcal (Infections and infestations) | 0 | 2 | 0
Accidental exposure to product (Injury, poisoning and procedural complications) | 0 | 1 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 2 | 0 | 2
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 2 | 2
Anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 10 | 5 | 9
Arterial injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Back injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Brain contusion (Injury, poisoning and procedural complications) | 2 | 0 | 1
Burns second degree (Injury, poisoning and procedural complications) | 1 | 0 | 0
Burns third degree (Injury, poisoning and procedural complications) | 0 | 0 | 1
Cartilage injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 4 | 0 | 5
Chest injury (Injury, poisoning and procedural complications) | 1 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 3
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 2
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 2 | 4
Delayed spinal fusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Eye contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 4 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 8 | 11 | 10
Fat embolism (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 4 | 3 | 3
Femur fracture (Injury, poisoning and procedural complications) | 11 | 7 | 18
Fibula fracture (Injury, poisoning and procedural complications) | 3 | 0 | 2
Foetal exposure during pregnancy (Injury, poisoning and procedural complications) | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Foreign body (Injury, poisoning and procedural complications) | 0 | 0 | 1
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 2 | 0
Heat exhaustion (Injury, poisoning and procedural complications) | 2 | 1 | 0
Hepatic rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 8 | 11 | 16
Humerus fracture (Injury, poisoning and procedural complications) | 4 | 5 | 5
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Intervertebral disc injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 6 | 5 | 3
Joint injury (Injury, poisoning and procedural complications) | 1 | 1 | 2
Laceration (Injury, poisoning and procedural complications) | 3 | 1 | 0
Ligament injury (Injury, poisoning and procedural complications) | 0 | 0 | 2
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 4 | 0
Limb crushing injury (Injury, poisoning and procedural complications) | 0 | 2 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 3 | 2 | 3
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 4 | 3
Multiple fractures (Injury, poisoning and procedural complications) | 2 | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 2 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Nerve injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 3 | 3
Patella fracture (Injury, poisoning and procedural complications) | 0 | 4 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Perirenal haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post concussion syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 2 | 0 | 2
Post procedural constipation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 3 | 3 | 3
Post procedural oedema (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural swelling (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 0 | 1
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 1 | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 2 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 3 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Radius fracture (Injury, poisoning and procedural complications) | 9 | 1 | 0
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 4 | 5 | 8
Road traffic accident (Injury, poisoning and procedural complications) | 4 | 9 | 6
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 | 0 | 10
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 4
Spinal shock (Injury, poisoning and procedural complications) | 1 | 0 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0 | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 6 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 4 | 6 | 2
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 2
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 6
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 2 | 4
Traumatic arthritis (Injury, poisoning and procedural complications) | 0 | 0 | 1
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 | 1 | 0
Traumatic renal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 2 | 2 | 4
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 1
Urostomy complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 | 1 | 0
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 3
Wound decomposition (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 1
Wound necrosis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound secretion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 4 | 2 | 3
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Aspiration bronchial (Investigations) | 0 | 1 | 0
Biopsy anus (Investigations) | 0 | 0 | 1
Biopsy breast (Investigations) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1
Blood chromium increased (Investigations) | 0 | 0 | 1
Blood creatine abnormal (Investigations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 3
Blood glucose abnormal (Investigations) | 0 | 0 | 1
Blood glucose increased (Investigations) | 1 | 0 | 0
Blood iron decreased (Investigations) | 0 | 1 | 0
Blood pressure increased (Investigations) | 1 | 2 | 3
Blood pressure systolic increased (Investigations) | 0 | 0 | 1
Blood triglycerides increased (Investigations) | 0 | 1 | 0
Clostridium test positive (Investigations) | 0 | 2 | 0
Ejection fraction (Investigations) | 1 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 1 | 0
Electrocardiogram abnormal (Investigations) | 0 | 0 | 2
Endoscopy gastrointestinal (Investigations) | 0 | 1 | 0
Fibrin D dimer increased (Investigations) | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1
Heart rate irregular (Investigations) | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 2 | 0 | 1
Liver function test increased (Investigations) | 0 | 0 | 1
Occult blood positive (Investigations) | 1 | 0 | 0
Oxygen saturation decreased (Investigations) | 1 | 0 | 1
Platelet count decreased (Investigations) | 0 | 1 | 0
Platelet function test abnormal (Investigations) | 0 | 1 | 0
Staphylococcus test positive (Investigations) | 0 | 0 | 1
Transaminases increased (Investigations) | 2 | 0 | 1
Troponin increased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 10 | 20 | 13
Diabetes mellitus (Metabolism and nutrition disorders) | 5 | 2 | 6
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 | 1 | 4
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 4 | 4
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 2 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1 | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 3 | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 4 | 2
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperosmolar hyperglycaemic state (Metabolism and nutrition disorders) | 2 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 6 | 7 | 8
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 9 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 7 | 8 | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 3 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 2 | 1
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 1
Obesity (Metabolism and nutrition disorders) | 5 | 5 | 5
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 44 | 33 | 39
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 17 | 20
Bone cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bone disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bone erosion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 8 | 7 | 2
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Felty's syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Fracture malunion (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 7 | 13 | 11
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 3 | 0 | 5
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 19 | 16 | 16
Joint ankylosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint instability (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Knee deformity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Kyphosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 13 | 15 | 20
Meniscal degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 31 | 33 | 32
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 7
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 5 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 5 | 3 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 201 | 206 | 189
Osteoarthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 7 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Polymyositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 3 | 4 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 8 | 5 | 3
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 10 | 7 | 10
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 13 | 12 | 7
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 16 | 4
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 7 | 7 | 10
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Vertebral osteophyte (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 1
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 8 | 4
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3 | 2
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 20 | 11 | 10
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Breast cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bronchioloalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Carcinoid tumour of the duodenum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Carcinoid tumour of the small bowel (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Carcinoid tumour of the stomach (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 2
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Colon cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Diffuse large B-cell lymphoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 4
Endometrial cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Endometrial cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Female reproductive neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Follicle centre lymphoma, follicular grade I, II, III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastrointestinal melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Gastrointestinal stromal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Hairy cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Head and neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3 | 5
Large cell lung cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Lip neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lobular breast carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 1
Lung adenocarcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Lung carcinoma cell type unspecified stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 | 7 | 12
Lung squamous cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
Malignant mediastinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1 | 3
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Non-Hodgkin's lymphoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 1
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Ovarian cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 7 | 3
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Pancreatic carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancreatic carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Paraproteinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Parathyroid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 3
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 19 | 20
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4 | 2
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 2
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Sweat gland tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 1
Transitional cell cancer of the renal pelvis and ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
Triple negative breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 5 | 3
Altered state of consciousness (Nervous system disorders) | 0 | 1 | 0
Amnesia (Nervous system disorders) | 0 | 1 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 1
Autonomic neuropathy (Nervous system disorders) | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 1
Basal ganglia infarction (Nervous system disorders) | 0 | 1 | 0
Basal ganglia stroke (Nervous system disorders) | 0 | 0 | 1
Brachial plexopathy (Nervous system disorders) | 0 | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 0 | 1
Carotid arteriosclerosis (Nervous system disorders) | 1 | 0 | 0
Carotid artery disease (Nervous system disorders) | 0 | 0 | 1
Carotid artery dissection (Nervous system disorders) | 1 | 0 | 0
Carotid artery occlusion (Nervous system disorders) | 2 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 5 | 5 | 3
Carotid artery thrombosis (Nervous system disorders) | 1 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 2 | 2 | 1
Central nervous system lesion (Nervous system disorders) | 0 | 0 | 1
Central-alveolar hypoventilation (Nervous system disorders) | 0 | 0 | 1
Cerebellar infarction (Nervous system disorders) | 0 | 1 | 1
Cerebral cyst (Nervous system disorders) | 0 | 1 | 0
Cerebral haematoma (Nervous system disorders) | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 4 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 2
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 39 | 34 | 34
Cerebrovascular disorder (Nervous system disorders) | 1 | 0 | 1
Cervical cord compression (Nervous system disorders) | 1 | 0 | 0
Cervical myelopathy (Nervous system disorders) | 3 | 1 | 1
Cervical radiculopathy (Nervous system disorders) | 1 | 5 | 2
Chorea (Nervous system disorders) | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0
Complex regional pain syndrome (Nervous system disorders) | 1 | 0 | 0
Dementia (Nervous system disorders) | 2 | 1 | 1
Dementia Alzheimer's type (Nervous system disorders) | 0 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1
Diabetic hyperosmolar coma (Nervous system disorders) | 2 | 0 | 0
Diabetic neuropathy (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 6 | 5 | 6
Dural arteriovenous fistula (Nervous system disorders) | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 2 | 0 | 3
Dyskinesia (Nervous system disorders) | 0 | 0 | 1
Embolic stroke (Nervous system disorders) | 0 | 0 | 1
Encephalomalacia (Nervous system disorders) | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1 | 3
Epidural lipomatosis (Nervous system disorders) | 1 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 0 | 1
Facial paralysis (Nervous system disorders) | 1 | 2 | 2
Facial paresis (Nervous system disorders) | 0 | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 2
Headache (Nervous system disorders) | 4 | 6 | 0
Hemiparesis (Nervous system disorders) | 0 | 1 | 1
Hydrocephalus (Nervous system disorders) | 0 | 1 | 0
Hypertensive encephalopathy (Nervous system disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 2 | 4 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 1 | 0
IIIrd nerve paralysis (Nervous system disorders) | 1 | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 1 | 4 | 3
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 2 | 3 | 8
Lacunar infarction (Nervous system disorders) | 1 | 2 | 1
Lacunar stroke (Nervous system disorders) | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 6 | 1 | 1
Lumbar radiculopathy (Nervous system disorders) | 1 | 4 | 3
Mental impairment (Nervous system disorders) | 1 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 2 | 0 | 1
Migraine (Nervous system disorders) | 5 | 2 | 1
Migraine with aura (Nervous system disorders) | 1 | 0 | 0
Monoparesis (Nervous system disorders) | 0 | 0 | 1
Multiple sclerosis relapse (Nervous system disorders) | 1 | 0 | 0
Myelopathy (Nervous system disorders) | 0 | 0 | 1
Nerve compression (Nervous system disorders) | 0 | 1 | 2
Nerve root compression (Nervous system disorders) | 1 | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 1
Neurological symptom (Nervous system disorders) | 1 | 0 | 0
Neuromyopathy (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0
Normal pressure hydrocephalus (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 2 | 2
Paraplegia (Nervous system disorders) | 0 | 0 | 1
Parkinsonism (Nervous system disorders) | 0 | 0 | 1
Presyncope (Nervous system disorders) | 2 | 6 | 4
Quadriparesis (Nervous system disorders) | 0 | 0 | 1
Quadriplegia (Nervous system disorders) | 1 | 0 | 0
Radial nerve palsy (Nervous system disorders) | 0 | 0 | 1
Radicular pain (Nervous system disorders) | 0 | 0 | 2
Radiculopathy (Nervous system disorders) | 1 | 3 | 0
Sacral radiculopathy (Nervous system disorders) | 0 | 0 | 1
Sciatica (Nervous system disorders) | 1 | 2 | 2
Seizure (Nervous system disorders) | 6 | 8 | 4
Senile dementia (Nervous system disorders) | 0 | 1 | 0
Spinal claudication (Nervous system disorders) | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 2
Spondylitic myelopathy (Nervous system disorders) | 1 | 2 | 1
Status epilepticus (Nervous system disorders) | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 3 | 2 | 1
Syncope (Nervous system disorders) | 19 | 21 | 31
Thalamic infarction (Nervous system disorders) | 0 | 0 | 2
Toxic encephalopathy (Nervous system disorders) | 1 | 0 | 1
Transient global amnesia (Nervous system disorders) | 1 | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 22 | 29 | 28
Tremor (Nervous system disorders) | 1 | 0 | 1
Trigeminal neuralgia (Nervous system disorders) | 1 | 1 | 0
Unresponsive to stimuli (Nervous system disorders) | 0 | 0 | 1
Vascular encephalopathy (Nervous system disorders) | 1 | 0 | 2
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Device breakage (Product Issues) | 0 | 0 | 1
Device connection issue (Product Issues) | 1 | 0 | 0
Device dislocation (Product Issues) | 1 | 1 | 4
Device failure (Product Issues) | 1 | 1 | 4
Device loosening (Product Issues) | 0 | 0 | 1
Device malfunction (Product Issues) | 0 | 0 | 1
Device material issue (Product Issues) | 1 | 0 | 0
Lead dislodgement (Product Issues) | 1 | 0 | 0
Stent malfunction (Product Issues) | 1 | 0 | 0
Acute psychosis (Psychiatric disorders) | 0 | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 4
Bipolar I disorder (Psychiatric disorders) | 0 | 1 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 1
Confusional state (Psychiatric disorders) | 3 | 2 | 1
Delirium (Psychiatric disorders) | 0 | 1 | 4
Depression (Psychiatric disorders) | 3 | 5 | 3
Depression suicidal (Psychiatric disorders) | 1 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 1
Drug abuse (Psychiatric disorders) | 0 | 1 | 0
Dysphoria (Psychiatric disorders) | 0 | 0 | 1
Hallucination, auditory (Psychiatric disorders) | 0 | 0 | 1
Hypomania (Psychiatric disorders) | 0 | 0 | 1
Major depression (Psychiatric disorders) | 2 | 2 | 3
Mental status changes (Psychiatric disorders) | 10 | 5 | 8
Panic attack (Psychiatric disorders) | 0 | 1 | 2
Paranoia (Psychiatric disorders) | 0 | 0 | 1
Post-traumatic stress disorder (Psychiatric disorders) | 2 | 0 | 0
Schizoaffective disorder (Psychiatric disorders) | 0 | 1 | 2
Schizophrenia (Psychiatric disorders) | 1 | 2 | 2
Substance abuse (Psychiatric disorders) | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 4 | 4
Suicide attempt (Psychiatric disorders) | 2 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 36 | 39 | 31
Acute prerenal failure (Renal and urinary disorders) | 0 | 1 | 0
Bladder outlet obstruction (Renal and urinary disorders) | 0 | 0 | 1
Bladder prolapse (Renal and urinary disorders) | 2 | 3 | 1
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 1
Calculus bladder (Renal and urinary disorders) | 1 | 0 | 1
Calculus urethral (Renal and urinary disorders) | 0 | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 2 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0
Hypertensive nephropathy (Renal and urinary disorders) | 0 | 1 | 0
Incontinence (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 7 | 10 | 11
Nephropathy (Renal and urinary disorders) | 1 | 0 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 0 | 1
Renal artery stenosis (Renal and urinary disorders) | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 1
Renal cyst haemorrhage (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 7 | 21 | 18
Renal haematoma (Renal and urinary disorders) | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 2 | 2 | 1
Renal injury (Renal and urinary disorders) | 1 | 0 | 0
Renal mass (Renal and urinary disorders) | 1 | 1 | 0
Stag horn calculus (Renal and urinary disorders) | 0 | 0 | 1
Stress urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 2 | 3 | 1
Urethral stenosis (Renal and urinary disorders) | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 2
Urinary retention (Renal and urinary disorders) | 1 | 3 | 0
Urine flow decreased (Renal and urinary disorders) | 0 | 0 | 1
Adnexa uteri mass (Reproductive system and breast disorders) | 1 | 0 | 0
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 4 | 5 | 4
Breast disorder (Reproductive system and breast disorders) | 1 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 1 | 1 | 1
Colpocele (Reproductive system and breast disorders) | 0 | 1 | 0
Cystocele (Reproductive system and breast disorders) | 4 | 3 | 1
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 | 0 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 2
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 3 | 1 | 1
Ovarian mass (Reproductive system and breast disorders) | 0 | 1 | 0
Pelvic adhesions (Reproductive system and breast disorders) | 0 | 0 | 1
Pelvic floor muscle weakness (Reproductive system and breast disorders) | 1 | 0 | 1
Pelvic prolapse (Reproductive system and breast disorders) | 1 | 0 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0
Prostatic obstruction (Reproductive system and breast disorders) | 0 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0 | 1
Rectocele (Reproductive system and breast disorders) | 2 | 1 | 2
Spermatocele (Reproductive system and breast disorders) | 0 | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 1 | 1 | 1
Uterovaginal prolapse (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 4 | 2 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 | 11 | 4
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 9 | 13 | 10
Asthma-chronic obstructive pulmonary disease overlap syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 29 | 30 | 31
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 | 24 | 24
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 6
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 4
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 6
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 4
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 18 | 10 | 21
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 4
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 3
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 | 14 | 10
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Vocal cord inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 3 | 4 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 3 | 5 | 1
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Leukoplakia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Melanocytic hyperplasia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Panniculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash vesicular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 4 | 1
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Activities of daily living impaired (Social circumstances) | 0 | 1 | 0
Immobile (Social circumstances) | 1 | 0 | 0
Physical assault (Social circumstances) | 0 | 0 | 1
Bladder operation (Surgical and medical procedures) | 1 | 0 | 0
Cardiac pacemaker replacement (Surgical and medical procedures) | 0 | 0 | 1
Colporrhaphy (Surgical and medical procedures) | 0 | 1 | 0
Coronary arterial stent insertion (Surgical and medical procedures) | 1 | 0 | 0
Coronary revascularisation (Surgical and medical procedures) | 0 | 1 | 0
Cystocele repair (Surgical and medical procedures) | 1 | 0 | 0
Gastric banding (Surgical and medical procedures) | 0 | 0 | 1
Hernia repair (Surgical and medical procedures) | 0 | 0 | 1
Hip arthroplasty (Surgical and medical procedures) | 2 | 2 | 3
Hysterectomy (Surgical and medical procedures) | 0 | 1 | 0
Inguinal hernia repair (Surgical and medical procedures) | 1 | 0 | 0
Joint fluid drainage (Surgical and medical procedures) | 1 | 0 | 0
Knee arthroplasty (Surgical and medical procedures) | 1 | 1 | 3
Ligament operation (Surgical and medical procedures) | 0 | 1 | 0
Medical device removal (Surgical and medical procedures) | 0 | 0 | 1
Oophorectomy (Surgical and medical procedures) | 1 | 0 | 0
Parovarian cystectomy (Surgical and medical procedures) | 0 | 0 | 1
Renal artery stent placement (Surgical and medical procedures) | 1 | 0 | 0
Renal stone removal (Surgical and medical procedures) | 1 | 0 | 0
Shoulder arthroplasty (Surgical and medical procedures) | 0 | 2 | 2
Shoulder operation (Surgical and medical procedures) | 1 | 0 | 0
Spinal decompression (Surgical and medical procedures) | 0 | 2 | 0
Spinal fusion surgery (Surgical and medical procedures) | 0 | 1 | 1
Spinal operation (Surgical and medical procedures) | 1 | 0 | 1
Tenoplasty (Surgical and medical procedures) | 0 | 1 | 0
Thyroidectomy (Surgical and medical procedures) | 0 | 0 | 1
Vascular operation (Surgical and medical procedures) | 0 | 1 | 0
Wound drainage (Surgical and medical procedures) | 0 | 0 | 1
Accelerated hypertension (Vascular disorders) | 1 | 0 | 1
Aneurysm (Vascular disorders) | 0 | 0 | 2
Angiopathy (Vascular disorders) | 1 | 0 | 0
Aortic aneurysm (Vascular disorders) | 10 | 4 | 4
Aortic aneurysm rupture (Vascular disorders) | 0 | 1 | 1
Aortic arteriosclerosis (Vascular disorders) | 1 | 1 | 1
Aortic calcification (Vascular disorders) | 0 | 1 | 0
Aortic dilatation (Vascular disorders) | 0 | 0 | 2
Aortic dissection (Vascular disorders) | 1 | 0 | 0
Aortic stenosis (Vascular disorders) | 2 | 3 | 7
Arterial occlusive disease (Vascular disorders) | 1 | 2 | 2
Arteriosclerosis (Vascular disorders) | 1 | 2 | 3
Arteriovenous fistula (Vascular disorders) | 0 | 0 | 1
Bleeding varicose vein (Vascular disorders) | 0 | 0 | 2
Blue toe syndrome (Vascular disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 12 | 11 | 12
Extravasation blood (Vascular disorders) | 0 | 1 | 0
Extremity necrosis (Vascular disorders) | 3 | 1 | 0
Haematoma (Vascular disorders) | 2 | 1 | 4
Hypertension (Vascular disorders) | 18 | 35 | 21
Hypertensive crisis (Vascular disorders) | 4 | 7 | 14
Hypertensive emergency (Vascular disorders) | 1 | 2 | 2
Hypotension (Vascular disorders) | 7 | 13 | 9
Hypovolaemic shock (Vascular disorders) | 0 | 1 | 0
Intermittent claudication (Vascular disorders) | 2 | 1 | 0
Internal haemorrhage (Vascular disorders) | 0 | 0 | 1
Ischaemia (Vascular disorders) | 1 | 1 | 2
Labile hypertension (Vascular disorders) | 0 | 1 | 0
Leriche syndrome (Vascular disorders) | 0 | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 2
Malignant hypertension (Vascular disorders) | 1 | 2 | 3
Neurogenic shock (Vascular disorders) | 1 | 0 | 0
Orthostatic hypertension (Vascular disorders) | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 2 | 3 | 3
Arterial thrombosis (Vascular disorders) | 0 | 0 | 2
Penetrating aortic ulcer (Vascular disorders) | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 2 | 2 | 4
Peripheral artery aneurysm (Vascular disorders) | 0 | 2 | 0
Peripheral artery occlusion (Vascular disorders) | 2 | 3 | 1
Peripheral artery stenosis (Vascular disorders) | 1 | 0 | 2
Peripheral artery thrombosis (Vascular disorders) | 2 | 1 | 2
Peripheral ischaemia (Vascular disorders) | 3 | 2 | 0
Peripheral vascular disorder (Vascular disorders) | 4 | 3 | 5
Peripheral venous disease (Vascular disorders) | 0 | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0 | 2
Shock (Vascular disorders) | 2 | 0 | 0
Subclavian vein thrombosis (Vascular disorders) | 0 | 1 | 0
Systolic hypertension (Vascular disorders) | 0 | 1 | 1
Temporal arteritis (Vascular disorders) | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 2 | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 1 | 1 | 2
Thrombosis (Vascular disorders) | 3 | 2 | 1
Varicose vein (Vascular disorders) | 1 | 1 | 1
Vascular stenosis (Vascular disorders) | 0 | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 2 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 1
Bradycardia and atrial flutter with hospitalization cardiorespiratory arrest and ischemia dilated (Cardiac disorders) | 1 | 0 | 0 — Being Queried
Cardiomyopathy and non-ST elevation MI and atherosclerosis (Cardiac disorders) | 1 | 0 | 0 — Being Queried
Femoral popliteal occlusive disease (Vascular disorders) | 1 | 0 | 0 — Being Queried
Large granular lymphocyte (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 — Being Queried
Left hip surgical error (Surgical and medical procedures) | 1 | 0 | 0 — Being Queried
Metastatic hepatic adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 — Being Queried
Metastatic tumor possibly from squamous cell lung cancer and metastatic tumor cerebral tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 — Being Queried
MRSA (Infections and infestations) | 0 | 0 | 1 — Being Queried
Osteoarthritis with tibial component loosening (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 — Being Queried
Pyelonephritis with sepsis NFI (Infections and infestations) | 1 | 0 | 0 — Being Queried
Worsening osteoarthritis right hip replacement (Surgical and medical procedures) | 1 | 0 | 0 — Being Queried
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Celecoxib (N=8030) | Ibuprofen (N=7992) | Naproxen (N=7933)
Anaemia (Blood and lymphatic system disorders) | 207 | 405 | 310
Constipation (Gastrointestinal disorders) | 274 | 344 | 408
Diarrhoea (Gastrointestinal disorders) | 641 | 538 | 566
Dyspepsia (Gastrointestinal disorders) | 393 | 424 | 436
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 401 | 404 | 387
Nausea (Gastrointestinal disorders) | 425 | 482 | 502
Bronchitis (Infections and infestations) | 465 | 471 | 427
Sinusitis (Infections and infestations) | 373 | 421 | 375
Upper respiratory tract infection (Infections and infestations) | 584 | 595 | 560
Urinary tract infection (Infections and infestations) | 416 | 452 | 414
Arthralgia (Musculoskeletal and connective tissue disorders) | 764 | 659 | 764
Back pain (Musculoskeletal and connective tissue disorders) | 542 | 516 | 547
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 958 | 859 | 880
Pain in extremity (Musculoskeletal and connective tissue disorders) | 455 | 422 | 422
Headache (Nervous system disorders) | 361 | 409 | 365
Hypertension (Vascular disorders) | 762 | 1008 | 855

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.